CLINICAL TRIAL: NCT01035255
Title: A Multicenter, Randomized, Double-blind, Parallel Group, Active-controlled Study to Evaluate the Efficacy and Safety of LCZ696 Compared to Enalapril on Morbidity and Mortality in Patients With Chronic Heart Failure and Reduced Ejection Fraction
Brief Title: This Study Will Evaluate the Efficacy and Safety of LCZ696 Compared to Enalapril on Morbidity and Mortality of Patients With Chronic Heart Failure
Acronym: PARADIGM-HF
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Early termination was approved due to compelling efficacy of LCZ696 in patients with HF & reduced EF after final pre-specified interim analysis 28-Mar-2014.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLCZ696B2314; 2009-015834-31
Record Dates: First submitted 2009-12-16; First posted 2009-12-18 (Estimated); Results first posted 2015-09-07 (Estimated); Last update posted 2016-08-15 (Estimated); Status verified 2016-07

CONDITIONS: Heart Failure With Reduced Ejection Fraction
Keywords: chronic heart failure; cardiovascular death; hospitalization; outcome study; BNP; KCCQ; eGFR
MeSH Terms: interventions — sacubitril and valsartan sodium hydrate drug combination; BID protein, human; Enalapril

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- LCZ696 (Experimental): single-blind active run-in period consisted of treatment with enalapril 10 mg bid, followed by LCZ696 100 mg bid, and then LCZ696 200 mg bid over a total duration of 5 to 10 weeks. Temporary down-titration from LCZ696 200 mg bid to LCZ696 100 mg bid was allowed provided the patient was up-titrated back to LCZ696 200 mg bid and tolerated this dose for at least two weeks before being eligible for randomization. LCZ696 200mg BID during double blind treatment period
  Interventions: Drug: LCZ696 200 mg BID
- Enalapril (Active Comparator): single-blind active run-in period consisted of treatment with enalapril 10 mg bid, followed by LCZ696 100 mg bid, and then LCZ696 200 mg bid over a total duration of 5 to 10 weeks. Temporary down-titration from LCZ696 200 mg bid to LCZ696 100 mg bid was allowed provided the patient was up-titrated back to LCZ696 200 mg bid and tolerated this dose for at least two weeks before being eligible for randomization. Enalapril 10 mg BID during double blind treatment period
  Interventions: Drug: Enalapril 10 mg BID

INTERVENTIONS:
Drug: LCZ696 200 mg BID — LCZ696 200 mg BID
  Arms: LCZ696
Drug: Enalapril 10 mg BID — Enalapril 10 mg BID
  Arms: Enalapril

SUMMARY:
The study will evaluate the efficacy and safety of LCZ696 compared to enalapril on morbidity and mortality in patients with chronic heart failure (NYHA Class II - IV and EF =< 35%).

ELIGIBILITY:
Inclusion Criteria:

* Patients must give written informed consent before any assessment is performed.
* Outpatients ≥ 18 years of age, male or female.
* Patients with a diagnosis of CHF NYHA class II-IV and reduced ejection fraction (EF =< 35%) and elevated BNP.
* Patients must be on an ACEI or an ARB at a stable dose of at least enalapril 10 mg/d or equivalent for at least 4 weeks.
* Patients must be treated with a β-blocker, unless contraindicated or not tolerated, at a stable dose for at least 4 weeks.

Exclusion Criteria:

* Use of other investigational drugs at the time of enrollment, or within 30 days or 5 half-lives of enrollment, whichever is longer.
* History of hypersensitivity or allergy to any of the study drugs, drugs of similar chemical classes, ACEIs, ARBs, or NEP inhibitors as well as known or suspected contraindications to the study drugs.
* Previous history of intolerance to recommended target doses of ACEIs or ARBs
* Known history of angioedema.
* Requirement of treatment with both ACEIs and ARBs.
* Current acute decompensated HF (exacerbation of chronic HF manifested by signs and symptoms that may require intravenous therapy).
* Symptomatic hypotension and/or a SBP < 100 mmHg.
* Estimated GFR < 30 mL/min/1.73m2 as measured by the simplified MDRD formula
* Serum potassium > 5.2 mmol/L.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8442 (Actual)
Dates: Start 2009-12; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (791):
- United States (132):
  - Novartis Investigative Site, Birmingham, Alabama
  - Novartis Investigative Site, Huntsville, Alabama
  - Novartis Investigative Site, Mobile, Alabama
  - Novartis Investigative Site, Muscle Shoals, Alabama
  - Novartis Investigative Site, Anchorage, Alaska
  - Novartis Investigative Site, Gilbert, Arizona
  - Novartis Investigative Site, Phoenix, Arizona
  - Novartis Investigative Site, Little Rock, Arkansas
  - Novartis Investigative Site, Anaheim, California
  - Novartis Investigative Site, Bellflower, California
  - Novartis Investigative Site, Berkley, California
  - Novartis Investigative Site, Loma Linda, California
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, Mather, California
  - Novartis Investigative Site, Oceanside, California
  - Novartis Investigative Site, Palm Springs, California
  - Novartis Investigative Site, Pomona, California
  - Novartis Investigative Site, Sacramento, California
  - Novartis Investigative Site, San Diego, California
  - Novartis Investigative Site, Santa Rosa, California
  - Novartis Investigative Site, Stockton, California
  - Novartis Investigative Site, Tustin, California
  - Novartis Investigative Site, Denver, Colorado
  - Novartis Investigative Site, Stamford, Connecticut
  - Novartis Investigative Site, Washington D.C., District of Columbia
  - Novartis Investigative Site, Boynton Beach, Florida
  - Novartis Investigative Site, Davie, Florida
  - Novartis Investigative Site, Fort Lauderdale, Florida
  - Novartis Investigative Site, Gainesville, Florida
  - Novartis Investigative Site, Jacksonville, Florida
  - Novartis Investigative Site, Lakeland, Florida
  - Novartis Investigative Site, Leesburg, Florida
  - Novartis Investigative Site, Port Charlotte, Florida
  - Novartis Investigative Site, Tamarac, Florida
  - Novartis Investigative Site, Tampa, Florida
  - Novartis Investigative Site, Covington, Georgia
  - Novartis Investigative Site, Decatur, Georgia
  - Novartis Investigative Site, Honolulu, Hawaii
  - Novartis Investigative Site, Chicago, Illinois
  - Novartis Investigative Site, Maywood, Illinois
  - Novartis Investigative Site, Melrose Park, Illinois
  - Novartis Investigative Site, Park Ridge, Illinois
  - Novartis Investigative Site, Quincy, Illinois
  - Novartis Investigative Site, Des Moines, Iowa
  - Novartis Investigative Site, Pratt, Kansas
  - Novartis Investigative Site, Topeka, Kansas
  - Novartis Investigative Site, Wichita, Kansas
  - Novartis Investigative Site, Alexandria, Louisiana
  - Novartis Investigative Site, Covington, Louisiana
  - Novartis Investigative Site, Lafayette, Louisiana
  - Novartis Investigative Site, Slidell, Louisiana
  - Novartis Investigative Site, Biddeford, Maine
  - Novartis Investigative Site, South Portland, Maine
  - Novartis Investigative Site, Baltimore, Maryland
  - Novartis Investigative Site, Beltsville, Maryland
  - Novartis Investigative Site, Columbia, Maryland
  - Novartis Investigative Site, Nottingham, Maryland
  - Novartis Investigative Site, Ayer, Massachusetts
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Haverhill, Massachusetts
  - Novartis Investigative Site, Natick, Massachusetts
  - Novartis Investigative Site, Ann Arbor, Michigan
  - Novartis Investigative Site, Detroit, Michigan
  - Novartis Investigative Site, Lapeer, Michigan
  - Novartis Investigative Site, Saginaw, Michigan
  - Novartis Investigative Site, Minneapolis, Minnesota
  - Novartis Investigative Site, Saint Paul, Minnesota
  - Novartis Investigative Site, Picayune, Mississippi
  - Novartis Investigative Site, Rolling Fork, Mississippi
  - Novartis Investigative Site, Springfield, Missouri
  - Novartis Investigative Site, Fremont, Nebraska
  - Novartis Investigative Site, Grand Island, Nebraska
  - Novartis Investigative Site, Omaha, Nebraska
  - Novartis Investigative Site, Nashua, New Hampshire
  - Novartis Investigative Site, Elizabeth, New Jersey
  - Novartis Investigative Site, Hamilton, New Jersey
  - Novartis Investigative Site, New Brunswick, New Jersey
  - Novartis Investigative Site, Newark, New Jersey
  - Novartis Investigative Site, Ocean City, New Jersey
  - Novartis Investigative Site, Albuquerque, New Mexico
  - Novartis Investigative Site, Cordtlandt Manor, New York
  - Novartis Investigative Site, Laurelton, New York
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Northport, New York
  - Novartis Investigative Site, Asheboro, North Carolina
  - Novartis Investigative Site, Asheville, North Carolina
  - Novartis Investigative Site, Cary, North Carolina
  - Novartis Investigative Site, Greensboro, North Carolina
  - Novartis Investigative Site, Raleigh, North Carolina
  - Novartis Investigative Site, Wilmington, North Carolina
  - Novartis Investigative Site, Cadiz, Ohio
  - Novartis Investigative Site, Canton, Ohio
  - Novartis Investigative Site, Cincinnati, Ohio
  - Novartis Investigative Site, Cleveland, Ohio
  - Novartis Investigative Site, Columbus, Ohio
  - Novartis Investigative Site, Marion, Ohio
  - Novartis Investigative Site, Bartlesville, Oklahoma
  - Novartis Investigative Site, Oklahoma City, Oklahoma
  - Novartis Investigative Site, Stillwater, Oklahoma
  - Novartis Investigative Site, Tulsa, Oklahoma
  - Novartis Investigative Site, Portland, Oregon
  - Novartis Investigative Site, Aliquippa, Pennsylvania
  - Novartis Investigative Site, Beaver, Pennsylvania
  - Novartis Investigative Site, Philadelphia, Pennsylvania
  - Novartis Investigative Site, Pittsburgh, Pennsylvania
  - Novartis Investigative Site, Charleston, South Carolina
  - Novartis Investigative Site, Rapid City, South Dakota
  - Novartis Investigative Site, Memphis, Tennessee
  - Novartis Investigative Site, Nashville, Tennessee
  - Novartis Investigative Site, Amarillo, Texas
  - Novartis Investigative Site, Arlington, Texas
  - Novartis Investigative Site, Beaumont, Texas
  - Novartis Investigative Site, Brownsville, Texas
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Grapevine, Texas
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, Kingwood, Texas
  - Novartis Investigative Site, Livingston, Texas
  - Novartis Investigative Site, Lufkin, Texas
  - Novartis Investigative Site, Odessa, Texas
  - Novartis Investigative Site, Plano, Texas
  - Novartis Investigative Site, Tyler, Texas
  - Novartis Investigative Site, Layton, Utah
  - Novartis Investigative Site, Fredericksburg, Virginia
  - Novartis Investigative Site, Richmond, Virginia
  - Novartis Investigative Site, Seattle, Washington
  - Novartis Investigative Site, Spokane, Washington
  - Novartis Investigative Site, Tacoma, Washington
  - Novartis Investigative Site, Madison, Wisconsin
  - Novartis Investigative Site, Milwaukee, Wisconsin
  - Novartis Investigative Site, Waukesha, Wisconsin
  - Novartis Investigative Site, Wausau, Wisconsin
- Argentina (26):
  - Novartis Investigative Site, Buenos Aires, Buenos Aires
  - Novartis Investigative Site, Caba, Buenos Aires
  - Novartis Investigative Site, Ciudad Autonoma de Bs As, Buenos Aires
  - Novartis Investigative Site, Lanús, Buenos Aires
  - Novartis Investigative Site, Mar del Plata, Buenos Aires
  - Novartis Investigative Site, Munro, Buenos Aires
  - Novartis Investigative Site, Pilar, Buenos Aires
  - Novartis Investigative Site, Quilmes, Buenos Aires
  - Novartis Investigative Site, San Isidro, Buenos Aires
  - Novartis Investigative Site, Zárate, Buenos Aires
  - Novartis Investigative Site, Caba, Buenos Aires F.D.
  - Novartis Investigative Site, Trelew, Chubut Province
  - Novartis Investigative Site, Corrientes, Corrientes Province
  - Novartis Investigative Site, Córdoba, Córdoba Province
  - Novartis Investigative Site, Formosa, Formosa Province
  - Novartis Investigative Site, San Salvador de Jujuy, Jujuy Province
  - Novartis Investigative Site, Mendoza, Mendoza Province
  - Novartis Investigative Site, Cipolletti, Río Negro Province
  - Novartis Investigative Site, Salta, Salta Province
  - Novartis Investigative Site, Buenos Aires, San Juan Province
  - Novartis Investigative Site, San Juan, San Juan Province
  - Novartis Investigative Site, San Luis, San Luis Province
  - Novartis Investigative Site, Rosario, Santa Fe Province
  - Novartis Investigative Site, Santa Fe, Santa Fe Province
  - Novartis Investigative Site, Santiago del Estero, Santiago del Estero Province
  - Novartis Investigative Site, San Miguel de Tucumán, Tucumán Province
- Belgium (13):
  - Novartis Investigative Site, Heusden-Zolder, Belgium
  - Novartis Investigative Site, Antwerp
  - Novartis Investigative Site, Baudour
  - Novartis Investigative Site, Bonheiden
  - Novartis Investigative Site, Brasschaat
  - Novartis Investigative Site, Bruges
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Hasselt
  - Novartis Investigative Site, La Louvière
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Ottignies
  - Novartis Investigative Site, Ronse
- Brazil (19):
  - Novartis Investigative Site, Salvador, Estado de Bahia
  - Novartis Investigative Site, Brasília, Federal District
  - Novartis Investigative Site, Goiânia, Goiás
  - Novartis Investigative Site, São Luís, Maranhão
  - Novartis Investigative Site, Belo Horizonte, Minas Gerais
  - Novartis Investigative Site, Uberlândia, Minas Gerais
  - Novartis Investigative Site, Curitiba, Paraná
  - Novartis Investigative Site, Belém, Pará
  - Novartis Investigative Site, Recife, Pernambuco
  - Novartis Investigative Site, Rio de Janeiro, Rio de Janeiro
  - Novartis Investigative Site, Natal, Rio Grande do Norte
  - Novartis Investigative Site, Passo Fundo, Rio Grande do Sul
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, Marília, São Paulo
  - Novartis Investigative Site, Ribeirão Preto, São Paulo
  - Novartis Investigative Site, Santo André, São Paulo
  - Novartis Investigative Site, São José do Rio Preto, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
  - Novartis Investigative Site, Votuporanga, São Paulo
- Bulgaria (14):
  - Novartis Investigative Site, Burgas, Bulgaria
  - Novartis Investigative Site, Plovdiv, Bulgaria
  - Novartis Investigative Site, Sofia, Bulgaria
  - Novartis Investigative Site, Haskovo
  - Novartis Investigative Site, Pazardzhik
  - Novartis Investigative Site, Pleven
  - Novartis Investigative Site, Plovdiv
  - Novartis Investigative Site, Rousse
  - Novartis Investigative Site, Shumen
  - Novartis Investigative Site, Silistra
  - Novartis Investigative Site, Sofia
  - Novartis Investigative Site, Stara Zagora
  - Novartis Investigative Site, Varna
  - Novartis Investigative Site, Veliko Tarnovo
- Canada (23):
  - Novartis Investigative Site, New Westminster, British Columbia
  - Novartis Investigative Site, Surrey, British Columbia
  - Novartis Investigative Site, Victoria, British Columbia
  - Novartis Investigative Site, Moncton, New Brunswick
  - Novartis Investigative Site, Halifax, Nova Scotia
  - Novartis Investigative Site, Cambridge, Ontario
  - Novartis Investigative Site, Greater Sudbury, Ontario
  - Novartis Investigative Site, Kitchener, Ontario
  - Novartis Investigative Site, London, Ontario
  - Novartis Investigative Site, Oshawa, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Weston, Ontario
  - Novartis Investigative Site, Granby, Quebec
  - Novartis Investigative Site, Lachine, Quebec
  - Novartis Investigative Site, Laval, Quebec
  - Novartis Investigative Site, Lévis, Quebec
  - Novartis Investigative Site, Longueuil, Quebec
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Sainte-Foy, Quebec
  - Novartis Investigative Site, Sherbrooke, Quebec
  - Novartis Investigative Site, St-Georges Beauce, Quebec
  - Novartis Investigative Site, Thetford-Mines, Quebec
  - Novartis Investigative Site, Regina, Saskatchewan
- Chile (7):
  - Novartis Investigative Site, Los Ángeles, Bio Bio
  - Novartis Investigative Site, Temuco, Cautin
  - Novartis Investigative Site, Temuco, Región de la Araucanía
  - Novartis Investigative Site, San Miguel, Santiago Metropolitan
  - Novartis Investigative Site, Santiago, Santiago Metropolitan
  - Novartis Investigative Site, Vitacura, Santiago Metropolitan
  - Novartis Investigative Site, Talcahuano
- China (12):
  - Novartis Investigative Site, Beijing, Beijing Municipality
  - Novartis Investigative Site, Harbin, Heilongjiang
  - Novartis Investigative Site, Changsha, Hunan
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Shenyang, Liaoning
  - Novartis Investigative Site, Xi’an, Shanxi
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Baotou
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Chongqing
  - Novartis Investigative Site, Shanghai
- Colombia (12):
  - Novartis Investigative Site, Barranquilla, Atlántico
  - Novartis Investigative Site, Barranquilla, Colombia
  - Novartis Investigative Site, Cali, Colombia
  - Novartis Investigative Site, Cartegena, Colombia
  - Novartis Investigative Site, Bogota, Cundinamarca
  - Novartis Investigative Site, Cartagena, Departamento de Bolívar
  - Novartis Investigative Site, Bucaramanga, Santander Department
  - Novartis Investigative Site, Floridablanca, Santander Department
  - Novartis Investigative Site, Barranquilla
  - Novartis Investigative Site, Bogotá
  - Novartis Investigative Site, Florida Blanca
  - Novartis Investigative Site, Medellín
- Czechia (22):
  - Novartis Investigative Site, Beroun, Czech Republic
  - Novartis Investigative Site, Brandýs nad Labem, Czech Republic
  - Novartis Investigative Site, Hořovice, Czech Republic
  - Novartis Investigative Site, Jablonec nad Nisou, Czech Republic
  - Novartis Investigative Site, Karlovy Vary, Czech Republic
  - Novartis Investigative Site, Kladno, Czech Republic
  - Novartis Investigative Site, Klatovy, Czech Republic
  - Novartis Investigative Site, Liberec V Kristianova, Czech Republic
  - Novartis Investigative Site, Mělník, Czech Republic
  - Novartis Investigative Site, Olomouc, Czech Republic
  - Novartis Investigative Site, Pilsen, Czech Republic
  - Novartis Investigative Site, Prague, Czech Republic
  - Novartis Investigative Site, Prague 10, Vrsovice, Czech Republic
  - Novartis Investigative Site, Semily, Czech Republic
  - Novartis Investigative Site, Strakonice, Czech Republic
  - Novartis Investigative Site, Třebíč, Czech Republic
  - Novartis Investigative Site, Ústí nad Labem, Czech Republic
  - Novartis Investigative Site, Bílovec, CZE
  - Novartis Investigative Site, Prague, CZE
  - Novartis Investigative Site, Kolín
  - Novartis Investigative Site, Prague
  - Novartis Investigative Site, Uherské Hradiště
- Denmark (10):
  - Novartis Investigative Site, Hellerup, Denmark
  - Novartis Investigative Site, Aarhus C
  - Novartis Investigative Site, Copenhagen
  - Novartis Investigative Site, Esbjerg
  - Novartis Investigative Site, Herning
  - Novartis Investigative Site, Randers NØ
  - Novartis Investigative Site, Roskilde
  - Novartis Investigative Site, Svendborg
  - Novartis Investigative Site, Vejle
  - Novartis Investigative Site, Viborg
- Dominican Republic (2):
  - Novartis Investigative Site, Santo Domingo, Republica Dominicana
  - Novartis Investigative Site, Santo Domingo, Santo Domingo Province
- Ecuador (2):
  - Novartis Investigative Site, Guayaquil, Guayas
  - Novartis Investigative Site, Quito, Pichincha
- Estonia (4):
  - Novartis Investigative Site, Tallinn, Estonia
  - Novartis Investigative Site, Haabneeme, Viimsi Vald
  - Novartis Investigative Site, Tallinn
  - Novartis Investigative Site, Tartu
- Finland (5):
  - Novartis Investigative Site, Kuopio, Finland
  - Novartis Investigative Site, HUS
  - Novartis Investigative Site, Kemi
  - Novartis Investigative Site, Oulu
  - Novartis Investigative Site, Tampere
- France (26):
  - Novartis Investigative Site, Strasbourg, Cedex
  - Novartis Investigative Site, Abbeville
  - Novartis Investigative Site, Bayonne
  - Novartis Investigative Site, Béziers
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Caen
  - Novartis Investigative Site, Cholet
  - Novartis Investigative Site, Créteil
  - Novartis Investigative Site, Essey-lès-Nancy
  - Novartis Investigative Site, Grenoble
  - Novartis Investigative Site, Lagny-sur-Marne
  - Novartis Investigative Site, Langres
  - Novartis Investigative Site, Le Chesnay
  - Novartis Investigative Site, Le Plessis-Robinson
  - Novartis Investigative Site, Limoges
  - Novartis Investigative Site, Lomme
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Reims
  - Novartis Investigative Site, Rouen
  - Novartis Investigative Site, Saint-Aubin-lès-Elbeuf
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Tourcoing
  - Novartis Investigative Site, Valencienne
  - Novartis Investigative Site, Vandœuvre-lès-Nancy
- Germany (79):
  - Novartis Investigative Site, Mannheim, Baden-Wurttemberg
  - Novartis Investigative Site, Berlin, Germany
  - Novartis Investigative Site, Ludwigshafen, Germany
  - Novartis Investigative Site, Ahrensfelde
  - Novartis Investigative Site, Bad Homburg
  - Novartis Investigative Site, Bad Krozingen
  - Novartis Investigative Site, Bad Salzuflen
  - Novartis Investigative Site, Bad Schwartau
  - Novartis Investigative Site, Barsinghausen
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bernau
  - Novartis Investigative Site, Bitburg
  - Novartis Investigative Site, Bremen
  - Novartis Investigative Site, Buch
  - Novartis Investigative Site, Chemnitz
  - Novartis Investigative Site, Darmstadt
  - Novartis Investigative Site, Dessau
  - Novartis Investigative Site, Dietzenbach
  - Novartis Investigative Site, Dortmund
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Eilenburg
  - Novartis Investigative Site, Elsterwerda
  - Novartis Investigative Site, Erfurt
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Georgsmarienhütte
  - Novartis Investigative Site, Giengen an der Brenz
  - Novartis Investigative Site, Goch
  - Novartis Investigative Site, Graben-Neudorf
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hamminkeln
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Homburg
  - Novartis Investigative Site, Hoppegarten-Dahlwitz
  - Novartis Investigative Site, Huy / OT Anderbeck
  - Novartis Investigative Site, Ingelheim
  - Novartis Investigative Site, Jena
  - Novartis Investigative Site, Kallstadt
  - Novartis Investigative Site, Kassel
  - Novartis Investigative Site, Kelkheim
  - Novartis Investigative Site, Köthen
  - Novartis Investigative Site, Künzelsau
  - Novartis Investigative Site, Langen
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Löhne
  - Novartis Investigative Site, Ludwigshafen
  - Novartis Investigative Site, Lübeck
  - Novartis Investigative Site, Lütjenburg
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Mannheim
  - Novartis Investigative Site, Meissen
  - Novartis Investigative Site, Meißen
  - Novartis Investigative Site, Mönchengladbach
  - Novartis Investigative Site, Mühldorf
  - Novartis Investigative Site, Mühlheim
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Neunkirchen
  - Novartis Investigative Site, Nienburg
  - Novartis Investigative Site, Offenbach
  - Novartis Investigative Site, Oldenburg i.H.
  - Novartis Investigative Site, Osnabrück
  - Novartis Investigative Site, Papenburg
  - Novartis Investigative Site, Rhaunen
  - Novartis Investigative Site, Riesa
  - Novartis Investigative Site, Rodgau
  - Novartis Investigative Site, Saint Ingbert - Oberwuerzbach
  - Novartis Investigative Site, Schenklengsfeld
  - Novartis Investigative Site, Schkeuditz
  - Novartis Investigative Site, Schwäbisch Hall
  - Novartis Investigative Site, Unterschneidheim
  - Novartis Investigative Site, Wangen
  - Novartis Investigative Site, Wardenburg
  - Novartis Investigative Site, Weeze
  - Novartis Investigative Site, Wermsdorf
  - Novartis Investigative Site, Westhofen
  - Novartis Investigative Site, Wetzlar-Naunheim
  - Novartis Investigative Site, Weyhe
  - Novartis Investigative Site, Wolmirstedt
- Novartis Investigative Site, Guatemala City, Departamento de Guatemala, Guatemala
- Hong Kong (3):
  - Novartis Investigative Site, Hong Kong, Hong Kong
  - Novartis Investigative Site, Hong Kong
  - Novartis Investigative Site, Hong Kong SAR
- Hungary (19):
  - Novartis Investigative Site, Pécs, Baranya
  - Novartis Investigative Site, Budapest, Hungary
  - Novartis Investigative Site, Cegléd, Hungary
  - Novartis Investigative Site, Miskolc, Hungary
  - Novartis Investigative Site, Baja
  - Novartis Investigative Site, Balatonfüred
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Eger
  - Novartis Investigative Site, Hódmezővásárhely
  - Novartis Investigative Site, Kaposvár
  - Novartis Investigative Site, Nagykanizsa
  - Novartis Investigative Site, Nyiregyháza
  - Novartis Investigative Site, Pécs
  - Novartis Investigative Site, Sopron
  - Novartis Investigative Site, Szeged
  - Novartis Investigative Site, Szekszárd
  - Novartis Investigative Site, Székesfehérvár
  - Novartis Investigative Site, Zalaegerszeg
- Iceland (2):
  - Novartis Investigative Site, Kopavogur
  - Novartis Investigative Site, Reykjavik
- India (32):
  - Novartis Investigative Site, Guntur, Andhra Pradesh
  - Novartis Investigative Site, Hyderabad, Andhra Pradesh
  - Novartis Investigative Site, Tirupati, Andhra Pradesh
  - Novartis Investigative Site, Visakhapatnam, Andhra Pradesh
  - Novartis Investigative Site, Hyderabad, Andhra Pradesh, India
  - Novartis Investigative Site, Ahmedabad, Gujarat
  - Novartis Investigative Site, Anand, Gujarat
  - Novartis Investigative Site, Rajkot, Gujarat
  - Novartis Investigative Site, Surat, Gujarat
  - Novartis Investigative Site, Vadodara, Gujarat
  - Novartis Investigative Site, Gurgaon, Haryana
  - Novartis Investigative Site, Indore, India
  - Novartis Investigative Site, Bangalore, Karnataka
  - Novartis Investigative Site, Banglaore, Karnataka
  - Novartis Investigative Site, Mangalore, Karnataka
  - Novartis Investigative Site, Mysore, Karnataka
  - Novartis Investigative Site, Kochi, Kerala
  - Novartis Investigative Site, Trivandrum, Kerala
  - Novartis Investigative Site, Mumbai, Maharashtra
  - Novartis Investigative Site, Nagpur, Maharashtra
  - Novartis Investigative Site, Nashik, Maharashtra
  - Novartis Investigative Site, Pune, Maharashtra
  - Novartis Investigative Site, Delhi, National Capital Territory of Delhi
  - Novartis Investigative Site, Ludhiana, Punjab
  - Novartis Investigative Site, Bikaner, Rajasthan
  - Novartis Investigative Site, Jaipur, Rajasthan
  - Novartis Investigative Site, Kota, Rajasthan
  - Novartis Investigative Site, Chennai, Tamil Nadu
  - Novartis Investigative Site, Lucknow, Uttar Pradesh
  - Novartis Investigative Site, Varanasi, Uttar Pradesh
  - Novartis Investigative Site, Ahmedabad
  - Novartis Investigative Site, Hyderabad
- Israel (7):
  - Novartis Investigative Site, Safed, Israel
  - Novartis Investigative Site, Ashkelon
  - Novartis Investigative Site, Hadera
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Rehovot
- Italy (37):
  - Novartis Investigative Site, Aosta, AO
  - Novartis Investigative Site, Cortona, AR
  - Novartis Investigative Site, Bergamo, BG
  - Novartis Investigative Site, Seriate, BG
  - Novartis Investigative Site, Treviglio, BG
  - Novartis Investigative Site, San Pietro Vernotico, BR
  - Novartis Investigative Site, Bolzano, BZ
  - Novartis Investigative Site, Cosenza, CS
  - Novartis Investigative Site, Catanzaro, CZ
  - Novartis Investigative Site, Cona, FE
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Pozzilli, IS
  - Novartis Investigative Site, Lido di Camaiore, LU
  - Novartis Investigative Site, Monza, MB
  - Novartis Investigative Site, Milazzo, ME
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Modena, MO
  - Novartis Investigative Site, Piove di Sacco, PD
  - Novartis Investigative Site, Perugia, PG
  - Novartis Investigative Site, Pisa, PI
  - Novartis Investigative Site, Pescia, PT
  - Novartis Investigative Site, Casorate Primo, PV
  - Novartis Investigative Site, Pavia, PV
  - Novartis Investigative Site, Stradella, PV
  - Novartis Investigative Site, Albano Laziale, RM
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Battipaglia, SA
  - Novartis Investigative Site, Cava de' Tirreni, SA
  - Novartis Investigative Site, Salerno, SA
  - Novartis Investigative Site, Sassari, SS
  - Novartis Investigative Site, Thiesi, SS
  - Novartis Investigative Site, Palmanova, UD
  - Novartis Investigative Site, San Daniele del Friuli, UD
  - Novartis Investigative Site, Tradate, VA
  - Novartis Investigative Site, Varese, VA
  - Novartis Investigative Site, Vibo Valentia, VV
- Latvia (6):
  - Novartis Investigative Site, Liepāja, LV
  - Novartis Investigative Site, Daugavplis
  - Novartis Investigative Site, Kuldīga
  - Novartis Investigative Site, Preiļi
  - Novartis Investigative Site, Riga
  - Novartis Investigative Site, Ventspils
- Lithuania (4):
  - Novartis Investigative Site, Kaunas
  - Novartis Investigative Site, Kėdainiai
  - Novartis Investigative Site, Šiauliai
  - Novartis Investigative Site, Vilnius
- Malaysia (3):
  - Novartis Investigative Site, Pulau Pinang, Pulau Pinang
  - Novartis Investigative Site, Kuching, Sarawak
  - Novartis Investigative Site, Kuala Lumpur
- Mexico (8):
  - Novartis Investigative Site, Aguascalientes, Aguascalientes
  - Novartis Investigative Site, Guadalajara, Jalisco
  - Novartis Investigative Site, Zapopan, Jalisco
  - Novartis Investigative Site, Mexico City, Mexico City
  - Novartis Investigative Site, Monterrey, Nuevo León
  - Novartis Investigative Site, Querétaro City, Querétaro
  - Novartis Investigative Site, San Juan del Río, Querétaro
  - Novartis Investigative Site, San Luis Potosí City, San Luis Potosí
- Netherlands (22):
  - Novartis Investigative Site, Ede, Netherlands
  - Novartis Investigative Site, Eindhoven, Netherlands
  - Novartis Investigative Site, Hardenberg, Netherlands
  - Novartis Investigative Site, Harderwijk, Netherlands
  - Novartis Investigative Site, Oss, NL
  - Novartis Investigative Site, 's-Hertogenbosch
  - Novartis Investigative Site, Amersfoort
  - Novartis Investigative Site, Arnhem
  - Novartis Investigative Site, Blaricum
  - Novartis Investigative Site, Breda
  - Novartis Investigative Site, Delft
  - Novartis Investigative Site, Goes
  - Novartis Investigative Site, Gorinchem
  - Novartis Investigative Site, Heerenveen
  - Novartis Investigative Site, Hengelo
  - Novartis Investigative Site, Hoorn
  - Novartis Investigative Site, Maastricht
  - Novartis Investigative Site, Nijmegen
  - Novartis Investigative Site, Sneek
  - Novartis Investigative Site, The Hague
  - Novartis Investigative Site, Tilburg
  - Novartis Investigative Site, Veldhoven
- Novartis Investigative Site, Panama City, Provincia de Panamá, Panama
- Peru (8):
  - Novartis Investigative Site, Arequipa, Arequipa
  - Novartis Investigative Site, Bellavista, Lima region
  - Novartis Investigative Site, Jesus Maria, Lima region
  - Novartis Investigative Site, La Molina, Lima region
  - Novartis Investigative Site, Lima Cercado, Lima region
  - Novartis Investigative Site, San Borja, Lima region
  - Novartis Investigative Site, San Isidro, Lima region
  - Novartis Investigative Site, San Miguel, Lima region
- Philippines (9):
  - Novartis Investigative Site, Lipa City, Batangas
  - Novartis Investigative Site, Quezon City, Manila
  - Novartis Investigative Site, Quezon City, National Capital Region
  - Novartis Investigative Site, Bulacan, Philippines
  - Novartis Investigative Site, Manila, Philippines
  - Novartis Investigative Site, San Juan City, Philippines
  - Novartis Investigative Site, Manila
  - Novartis Investigative Site, Pasig
  - Novartis Investigative Site, Quezon City
- Poland (13):
  - Novartis Investigative Site, Bialystok
  - Novartis Investigative Site, Gdynia
  - Novartis Investigative Site, Gliwice
  - Novartis Investigative Site, Golub-Dobrzyń
  - Novartis Investigative Site, Katowice
  - Novartis Investigative Site, Krakow
  - Novartis Investigative Site, Kutno
  - Novartis Investigative Site, Lodz
  - Novartis Investigative Site, Lublin
  - Novartis Investigative Site, Oława
  - Novartis Investigative Site, Skierniewice
  - Novartis Investigative Site, Wroclaw
  - Novartis Investigative Site, Zabrze
- Portugal (9):
  - Novartis Investigative Site, Porto, Porto District
  - Novartis Investigative Site, Amadora, Portugal
  - Novartis Investigative Site, Covilha, Portugal
  - Novartis Investigative Site, Guimarães, Portugal
  - Novartis Investigative Site, Lisbon, Portugal
  - Novartis Investigative Site, Penafiel, Portugal
  - Novartis Investigative Site, Portalegre, Portugal
  - Novartis Investigative Site, Vila Real, Portuigal
  - Novartis Investigative Site, Setúbal
- Romania (14):
  - Novartis Investigative Site, Bucharest, District 1
  - Novartis Investigative Site, Bucharest, District 2
  - Novartis Investigative Site, Bucharest, District 5
  - Novartis Investigative Site, Craiova, Jud. Dolj
  - Novartis Investigative Site, Timișoara, Jud. Timis
  - Novartis Investigative Site, Craiova, Jud.Dolj
  - Novartis Investigative Site, Ploieşti, Jud.Prahova
  - Novartis Investigative Site, Arad, Romania
  - Novartis Investigative Site, Bucharest, Romania
  - Novartis Investigative Site, Deva, Romania
  - Novartis Investigative Site, Timișoara, Romania
  - Novartis Investigative Site, Bucharest
  - Novartis Investigative Site, Piteşti
  - Novartis Investigative Site, Timișoara
- Russia (32):
  - Novartis Investigative Site, Gatchina
  - Novartis Investigative Site, Ivanovo
  - Novartis Investigative Site, Izhevsk
  - Novartis Investigative Site, Kazan'
  - Novartis Investigative Site, Kemerovo
  - Novartis Investigative Site, Kirov
  - Novartis Investigative Site, Krasnodar
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, N.Novgorod
  - Novartis Investigative Site, Nizhny Novgorod
  - Novartis Investigative Site, Novosibirsk
  - Novartis Investigative Site, Novosibirsk-117
  - Novartis Investigative Site, Orenburg
  - Novartis Investigative Site, Penza
  - Novartis Investigative Site, Perm
  - Novartis Investigative Site, Petrozavodsk
  - Novartis Investigative Site, Rostov-on-Don
  - Novartis Investigative Site, S-Petersburg
  - Novartis Investigative Site, S.-Petersburg
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Samara
  - Novartis Investigative Site, Saratov
  - Novartis Investigative Site, Smolensk
  - Novartis Investigative Site, St-Peterburg
  - Novartis Investigative Site, Syktyvkar
  - Novartis Investigative Site, Tula
  - Novartis Investigative Site, Tver'
  - Novartis Investigative Site, Vladimir
  - Novartis Investigative Site, Volgograd
  - Novartis Investigative Site, Voronezh
  - Novartis Investigative Site, Yaroslavl
  - Novartis Investigative Site, Yekaterinburg
- Novartis Investigative Site, Singapore, Singapore, Singapore
- Slovakia (18):
  - Novartis Investigative Site, Bratislava, Slovak Republic
  - Novartis Investigative Site, Brezno, Slovak Republic
  - Novartis Investigative Site, Košice, Slovak Republic
  - Novartis Investigative Site, Levice, Slovak Republic
  - Novartis Investigative Site, Prešov, Slovak Republic
  - Novartis Investigative Site, Svidník, Slovak Republic
  - Novartis Investigative Site, Vranov nad Topľou, Slovak Republic
  - Novartis Investigative Site, Bratislava, Slovakia
  - Novartis Investigative Site, Dunajská Streda, Slovakia
  - Novartis Investigative Site, Košice, Slovakia
  - Novartis Investigative Site, Kráľovský Chlmec, Slovakia
  - Novartis Investigative Site, Levice, Slovakia
  - Novartis Investigative Site, Lučenec, Slovakia
  - Novartis Investigative Site, Martin, Slovakia
  - Novartis Investigative Site, Nitra, Slovakia
  - Novartis Investigative Site, Trnava, Slovakia
  - Novartis Investigative Site, Bratislava
  - Novartis Investigative Site, Dolný Kubín
- South Africa (21):
  - Novartis Investigative Site, Mthatha, Eastern Cape
  - Novartis Investigative Site, Bloemfontein, Free State
  - Novartis Investigative Site, Soweto, Gauteng
  - Novartis Investigative Site, Middelburg, Mpumalanga
  - Novartis Investigative Site, Paarl, Western Cape
  - Novartis Investigative Site, Somerset West, Western Cape
  - Novartis Investigative Site, Alberton
  - Novartis Investigative Site, Bloemfontein
  - Novartis Investigative Site, Breyten
  - Novartis Investigative Site, Brits
  - Novartis Investigative Site, Cape Town
  - Novartis Investigative Site, Durban
  - Novartis Investigative Site, East London
  - Novartis Investigative Site, eMkhomazi
  - Novartis Investigative Site, Gatesville
  - Novartis Investigative Site, Johannesburg
  - Novartis Investigative Site, Kempton Park
  - Novartis Investigative Site, Port Elizabeth
  - Novartis Investigative Site, Pretoria
  - Novartis Investigative Site, Witbank
  - Novartis Investigative Site, Worcester
- South Korea (8):
  - Novartis Investigative Site, Busan, Busan
  - Novartis Investigative Site, Wŏnju, Gangwon-do
  - Novartis Investigative Site, Gwangju, Gwangju
  - Novartis Investigative Site, Suwon, Gyeonggi-do
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Daegu
  - Novartis Investigative Site, Pusan
  - Novartis Investigative Site, Seoul
- Spain (19):
  - Novartis Investigative Site, Almería, Andalusia
  - Novartis Investigative Site, Marbella, Andalusia
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Mallorca, Balearic Islands
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Sant Joan Despí, Catalonia
  - Novartis Investigative Site, Mérida, Extremadura
  - Novartis Investigative Site, A Coruña, Galicia
  - Novartis Investigative Site, Ferrol, Galicia
  - Novartis Investigative Site, Santiago de Compostela, Galicia
  - Novartis Investigative Site, Vigo, Galicia
  - Novartis Investigative Site, Alcalá de Henares, Madrid
  - Novartis Investigative Site, Madrid, Madrid
  - Novartis Investigative Site, Majadahonda, Madrid
  - Novartis Investigative Site, Móstoles, Madrid
  - Novartis Investigative Site, El Palmar, Murcia
  - Novartis Investigative Site, Alicante, Valencia
  - Novartis Investigative Site, Valencia, Valencia
- Sweden (8):
  - Novartis Investigative Site, Gothenburg
  - Novartis Investigative Site, Härnösand
  - Novartis Investigative Site, Helsingborg
  - Novartis Investigative Site, Karlshamn
  - Novartis Investigative Site, Lund
  - Novartis Investigative Site, Motala
  - Novartis Investigative Site, Stockholm
  - Novartis Investigative Site, Vällingby
- Taiwan (7):
  - Novartis Investigative Site, Taichung, Taiwan
  - Novartis Investigative Site, Taipei, Taiwan
  - Novartis Investigative Site, Tainan, Taiwan ROC
  - Novartis Investigative Site, Taipei, Taiwan, ROC
  - Novartis Investigative Site, Changhua
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Yilan
- Thailand (5):
  - Novartis Investigative Site, Taladkwan, Changwat Nonthaburi
  - Novartis Investigative Site, Muang, Muang
  - Novartis Investigative Site, Muang, Thailand
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Khon Kaen
- Turkey (Türkiye) (14):
  - Novartis Investigative Site, Istanbul, Turkey
  - Novartis Investigative Site, Izmir, Turkey
  - Novartis Investigative Site, Adana
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Antalya
  - Novartis Investigative Site, Balcova / Izmir
  - Novartis Investigative Site, Edirne
  - Novartis Investigative Site, Etlik / Ankara
  - Novartis Investigative Site, Haseki / Istanbul
  - Novartis Investigative Site, Istanbul
  - Novartis Investigative Site, Kocaeli
  - Novartis Investigative Site, Mersin
  - Novartis Investigative Site, Meselik / Eskisehir
  - Novartis Investigative Site, Sivas
- United Kingdom (48):
  - Novartis Investigative Site, Bristol, Bs2 8hw
  - Novartis Investigative Site, Cambridge, Cambrigdeshire
  - Novartis Investigative Site, Durham, County Durham
  - Novartis Investigative Site, Dorchester, Dorset
  - Novartis Investigative Site, Brighton, East Sussex
  - Novartis Investigative Site, Swansea, England
  - Novartis Investigative Site, Romford, Essex
  - Novartis Investigative Site, Basingstoke, Hampshire
  - Novartis Investigative Site, Portsmouth, Hampshire
  - Novartis Investigative Site, Royal Bridge Wells, Kent
  - Novartis Investigative Site, Oldham, Lancashire
  - Novartis Investigative Site, Leicester, Leicestershire
  - Novartis Investigative Site, Craigavon, Northern Ireland
  - Novartis Investigative Site, Dundee, Perthshire
  - Novartis Investigative Site, Taunton, Somerset
  - Novartis Investigative Site, Yeovil, Somerset
  - Novartis Investigative Site, Sheffield, South Yorkshire
  - Novartis Investigative Site, Redhill, Surrey
  - Novartis Investigative Site, South Shields, Tyne and Wear
  - Novartis Investigative Site, Dudley, West Midlands
  - Novartis Investigative Site, Sutton Coldfield, West Midlands
  - Novartis Investigative Site, Birmingham
  - Novartis Investigative Site, Blackpool
  - Novartis Investigative Site, Bournemouth
  - Novartis Investigative Site, Bradford
  - Novartis Investigative Site, Cheshire
  - Novartis Investigative Site, Coventry
  - Novartis Investigative Site, Croydon
  - Novartis Investigative Site, Darlington
  - Novartis Investigative Site, Exeter
  - Novartis Investigative Site, Inverness
  - Novartis Investigative Site, Kent
  - Novartis Investigative Site, Liverpool
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Londonderry
  - Novartis Investigative Site, Manchester
  - Novartis Investigative Site, Middlesbrough
  - Novartis Investigative Site, Milton Keynes
  - Novartis Investigative Site, Newport
  - Novartis Investigative Site, Norwich
  - Novartis Investigative Site, Poole
  - Novartis Investigative Site, Rotherham
  - Novartis Investigative Site, Stevenage
  - Novartis Investigative Site, Sunderland
  - Novartis Investigative Site, Surrey
  - Novartis Investigative Site, Vale of Glamorgan
  - Novartis Investigative Site, Worcester
  - Novartis Investigative Site, York
- Venezuela (4):
  - Novartis Investigative Site, Caracas, Distrito Federal
  - Novartis Investigative Site, Caracas, Miranda
  - Novartis Investigative Site, Maturín, Monagas
  - Novartis Investigative Site, Maracaibo, Zulia

REFERENCES:
- [Derived] Yang M, Henderson AD, Anand IS, Desai AS, Lam CSP, Maggioni AP, Martinez FA, Rouleau JL, Swedberg K, Vaduganathan M, van Veldhuisen DJ, Zannad F, Zile MR, Packer M, Rizkala A, Lewis EF, Jhund PS, Solomon SD, McMurray JJV. Sacubitril/valsartan and quality of life assessed using the EuroQol Five-dimension Three-level questionnaire level sum score (EQ-5D-3L-LSS) in patients with HFrEF and HFmrEF/HFpEF. Eur Heart J Cardiovasc Pharmacother. 2025 Nov 4;11(7):574-589. doi: 10.1093/ehjcvp/pvaf064. PMID 40839760
- [Derived] Chimura M, Butt JH, Matsumoto S, McMurray EGM, Henderson AD, Talebi A, Desai AS, Lefkowitz MP, Rizkala AR, Rouleau JL, Solomon SD, Swedberg K, Zile MR, Packer M, Jhund PS, McMurray JJV. Comprehensive Analysis of the Effects of Sacubitril/Valsartan According to Sex Among Patients With Heart Failure and Reduced Ejection Fraction in PARADIGM-HF. J Am Heart Assoc. 2025 May 6;14(9):e038249. doi: 10.1161/JAHA.124.038249. Epub 2025 Apr 23. PMID 40265590
- [Derived] Gupta SD, Butt JH, McMurray EGM, Talebi A, Matsumoto S, Rizkala AR, Henderson AD, Desai AS, Lefkowitz M, Packer M, Rouleau JL, Solomon SD, Swedberg K, Zile MR, Jhund PS, McMurray JJV; PARADIGM-HF Investigators and Committees. Effects of sacubitril/valsartan according to background beta-blocker therapy in patients with heart failure and reduced ejection fraction: Insights from PARADIGM-HF. Eur J Heart Fail. 2025 May;27(5):779-787. doi: 10.1002/ejhf.3515. Epub 2024 Nov 19. PMID 39563094
- [Derived] Lu H, Claggett BL, Packer M, Pfeffer MA, Swedberg K, Rouleau J, Zile MR, Lefkowitz M, Desai AS, Jhund PS, McMurray JJV, Solomon SD, Vaduganathan M. Visit-to-visit changes in heart rate in heart failure: A pooled participant-level analysis of the PARADIGM-HF and PARAGON-HF trials. Eur J Heart Fail. 2025 Jan;27(1):60-68. doi: 10.1002/ejhf.3487. Epub 2024 Oct 22. PMID 39439294
- [Derived] Lu H, Claggett BL, Packer M, Lam CSP, Swedberg K, Rouleau J, Zile MR, Lefkowitz M, Desai AS, Jhund P, McMurray JJV, Solomon SD, Vaduganathan M. Effects of Sacubitril/Valsartan on All-Cause Hospitalizations in Heart Failure: Post Hoc Analysis of the PARADIGM-HF and PARAGON-HF Randomized Clinical Trials. JAMA Cardiol. 2024 Nov 1;9(11):1047-1052. doi: 10.1001/jamacardio.2024.2566. PMID 39210725
- [Derived] Patel-Murray NL, Zhang L, Claggett BL, Xu D, Serrano-Fernandez P, Healey M, Wandel S, Chen CW, Jacob J, Xu H, Turner GM, Chutkow W, Yates DP, O'Donnell CJ, Prescott MF, Lefkowitz M, Gimpelewicz CR, Beste MT, Zhao F, Gou L, Desai AS, Jhund PS, Packer M, Pfeffer MA, Redfield MM, Rouleau JL, Zannad F, Zile MR, McMurray JJV, Mendelson MM, Solomon SD, Cunningham JW. Aptamer Proteomics for Biomarker Discovery in Heart Failure With Preserved Ejection Fraction: The PARAGON-HF Proteomic Substudy. J Am Heart Assoc. 2024 Jul 2;13(13):e033544. doi: 10.1161/JAHA.123.033544. Epub 2024 Jun 21. PMID 38904251
- [Derived] Chatur S, Neuen BL, Claggett BL, Beldhuis IE, Mc Causland FR, Desai AS, Rouleau JL, Zile MR, Lefkowitz MP, Packer M, McMurray JJV, Solomon SD, Vaduganathan M. Effects of Sacubitril/Valsartan Across the Spectrum of Renal Impairment in Patients With Heart Failure. J Am Coll Cardiol. 2024 Jun 4;83(22):2148-2159. doi: 10.1016/j.jacc.2024.03.392. Epub 2024 Apr 6. PMID 38588927
- [Derived] Bhatt AS, Vaduganathan M, Claggett BL, Kulac IJ, Anand IS, Desai AS, Fang JC, Hernandez AF, Jhund PS, Kosiborod MN, Sabatine MS, Shah SJ, Vardeny O, McMurray JJV, Solomon SD, Gaziano TA. Cost Effectiveness of Dapagliflozin for Heart Failure Across the Spectrum of Ejection Fraction: An Economic Evaluation Based on Pooled, Individual Participant Data From the DELIVER and DAPA-HF Trials. J Am Heart Assoc. 2024 Mar 5;13(5):e032279. doi: 10.1161/JAHA.123.032279. Epub 2024 Feb 23. PMID 38390793
- [Derived] Curtain JP, Adamson C, Docherty KF, Jhund PS, Desai AS, Lefkowitz MP, Rizkala AR, Rouleau JL, Swedberg K, Zile MR, Solomon SD, Packer M, McMurray JJV. Prevalent and Incident Anemia in PARADIGM-HF and the Effect of Sacubitril/Valsartan. JACC Heart Fail. 2023 Jul;11(7):749-759. doi: 10.1016/j.jchf.2022.12.012. Epub 2023 Apr 12. PMID 37407154
- [Derived] Kondo T, Dewan P, Anand IS, Desai AS, Packer M, Zile MR, Pfeffer MA, Solomon SD, Abraham WT, Shah SJ, Lam CSP, Jhund PS, McMurray JJV. Clinical Characteristics and Outcomes in Patients With Heart Failure: Are There Thresholds and Inflection Points in Left Ventricular Ejection Fraction and Thresholds Justifying a Clinical Classification? Circulation. 2023 Aug 29;148(9):732-749. doi: 10.1161/CIRCULATIONAHA.122.063642. Epub 2023 Jun 27. PMID 37366061
- [Derived] Tolomeo P, Butt JH, Kondo T, Campo G, Desai AS, Jhund PS, Kober L, Lefkowitz MP, Rouleau JL, Solomon SD, Swedberg K, Vaduganathan M, Zile MR, Packer M, McMurray JJV. Importance of cystatin C in estimating glomerular filtration rate: the PARADIGM-HF trial. Eur Heart J. 2023 Jun 25;44(24):2202-2212. doi: 10.1093/eurheartj/ehad210. PMID 37051752
- [Derived] Butt JH, Ibrahim W, Dewan P, Desai AS, Kober L, Prescott MF, Lefkowitz MP, Rouleau JL, Solomon SD, Zile MR, Packer M, Jhund PS, McMurray JJV. Urinary cGMP (Cyclic Guanosine Monophosphate)/BNP (B-Type Natriuretic Peptide) Ratio, Sacubitril/Valsartan, and Outcomes in Heart Failure With Reduced Ejection Fraction: An Analysis of the PARADIGM-HF Trial. Circ Heart Fail. 2023 Mar;16(3):e010111. doi: 10.1161/CIRCHEARTFAILURE.122.010111. Epub 2023 Jan 25. PMID 36943907
- [Derived] Rohde LE, Zimerman A, Vaduganathan M, Claggett BL, Packer M, Desai AS, Zile M, Rouleau J, Swedberg K, Lefkowitz M, Shi V, McMurray JJV, Solomon SD. Associations Between New York Heart Association Classification, Objective Measures, and Long-term Prognosis in Mild Heart Failure: A Secondary Analysis of the PARADIGM-HF Trial. JAMA Cardiol. 2023 Feb 1;8(2):150-158. doi: 10.1001/jamacardio.2022.4427. PMID 36477809
- [Derived] Vaduganathan M, Claggett BL, McMurray JJV, Solomon SD. Health Status Trajectories Before and After Hospitalization for Heart Failure. Circulation. 2022 Jun 21;145(25):1872-1874. doi: 10.1161/CIRCULATIONAHA.122.059282. Epub 2022 May 21. No abstract available. PMID 35603665
- [Derived] Toenges G, Mutze T, Jahn-Eimermacher A. A comparison of semiparametric approaches to evaluate composite endpoints in heart failure trials. Stat Med. 2021 Nov 20;40(26):5702-5724. doi: 10.1002/sim.9149. Epub 2021 Jul 30. PMID 34327735
- [Derived] Shen L, Claggett BL, Jhund PS, Abraham WT, Desai AS, Dickstein K, Gong J, Kober LV, Lefkowitz MP, Rouleau JL, Shi VC, Swedberg K, Zile MR, Solomon SD, McMurray JJV. Development and external validation of prognostic models to predict sudden and pump-failure death in patients with HFrEF from PARADIGM-HF and ATMOSPHERE. Clin Res Cardiol. 2021 Aug;110(8):1334-1349. doi: 10.1007/s00392-021-01888-x. Epub 2021 Jun 8. PMID 34101002
- [Derived] Shen L, Jhund PS, Anand IS, Bhatt AS, Desai AS, Maggioni AP, Martinez FA, Pfeffer MA, Rizkala AR, Rouleau JL, Swedberg K, Vaduganathan M, Vardeny O, van Veldhuisen DJ, Zannad F, Zile MR, Packer M, Solomon SD, McMurray JJV. Incidence and Outcomes of Pneumonia in Patients With Heart Failure. J Am Coll Cardiol. 2021 Apr 27;77(16):1961-1973. doi: 10.1016/j.jacc.2021.03.001. PMID 33888245
- [Derived] Ehteshami-Afshar S, Mooney L, Dewan P, Desai AS, Lang NN, Lefkowitz MP, Petrie MC, Rizkala AR, Rouleau JL, Solomon SD, Swedberg K, Shi VC, Zile MR, Packer M, McMurray JJV, Jhund PS, Hawkins NM. Clinical Characteristics and Outcomes of Patients With Heart Failure With Reduced Ejection Fraction and Chronic Obstructive Pulmonary Disease: Insights From PARADIGM-HF. J Am Heart Assoc. 2021 Feb 16;10(4):e019238. doi: 10.1161/JAHA.120.019238. Epub 2021 Jan 30. PMID 33522249
- [Derived] Kristensen SL, Castagno D, Shen L, Jhund PS, Docherty KF, Rorth R, Abraham WT, Desai AS, Dickstein K, Rouleau JL, Zile MR, Swedberg K, Packer M, Solomon SD, Kober L, McMurray JJV; PARADIGM-HF and ATMOSPHERE Committees and Investigators.. Prevalence and incidence of intra-ventricular conduction delays and outcomes in patients with heart failure and reduced ejection fraction: insights from PARADIGM-HF and ATMOSPHERE. Eur J Heart Fail. 2020 Dec;22(12):2370-2379. doi: 10.1002/ejhf.1972. Epub 2020 Sep 14. PMID 32720404
- [Derived] Docherty KF, Shen L, Castagno D, Petrie MC, Abraham WT, Bohm M, Desai AS, Dickstein K, Kober LV, Packer M, Rouleau JL, Solomon SD, Swedberg K, Vazir A, Zile MR, Jhund PS, McMurray JJV. Relationship between heart rate and outcomes in patients in sinus rhythm or atrial fibrillation with heart failure and reduced ejection fraction. Eur J Heart Fail. 2020 Mar;22(3):528-538. doi: 10.1002/ejhf.1682. Epub 2019 Dec 17. PMID 31849164
- [Derived] Dewan P, Rorth R, Raparelli V, Campbell RT, Shen L, Jhund PS, Petrie MC, Anand IS, Carson PE, Desai AS, Granger CB, Kober L, Komajda M, McKelvie RS, O'Meara E, Pfeffer MA, Pitt B, Solomon SD, Swedberg K, Zile MR, McMurray JJV. Sex-Related Differences in Heart Failure With Preserved Ejection Fraction. Circ Heart Fail. 2019 Dec;12(12):e006539. doi: 10.1161/CIRCHEARTFAILURE.119.006539. Epub 2019 Dec 9. PMID 31813280
- [Derived] Solomon SD, Vaduganathan M, L Claggett B, Packer M, Zile M, Swedberg K, Rouleau J, A Pfeffer M, Desai A, Lund LH, Kober L, Anand I, Sweitzer N, Linssen G, Merkely B, Luis Arango J, Vinereanu D, Chen CH, Senni M, Sibulo A, Boytsov S, Shi V, Rizkala A, Lefkowitz M, McMurray JJV. Sacubitril/Valsartan Across the Spectrum of Ejection Fraction in Heart Failure. Circulation. 2020 Feb 4;141(5):352-361. doi: 10.1161/CIRCULATIONAHA.119.044586. Epub 2019 Nov 17. PMID 31736342
- [Derived] Selvaraj S, Claggett B, Pozzi A, McMurray JJV, Jhund PS, Packer M, Desai AS, Lewis EF, Vaduganathan M, Lefkowitz MP, Rouleau JL, Shi VC, Zile MR, Swedberg K, Solomon SD. Prognostic Implications of Congestion on Physical Examination Among Contemporary Patients With Heart Failure and Reduced Ejection Fraction: PARADIGM-HF. Circulation. 2019 Oct 22;140(17):1369-1379. doi: 10.1161/CIRCULATIONAHA.119.039920. Epub 2019 Sep 12. PMID 31510768
- [Derived] Chandra A, Vaduganathan M, Lewis EF, Claggett BL, Rizkala AR, Wang W, Lefkowitz MP, Shi VC, Anand IS, Ge J, Lam CSP, Maggioni AP, Martinez F, Packer M, Pfeffer MA, Pieske B, Redfield MM, Rouleau JL, Van Veldhuisen DJ, Zannad F, Zile MR, McMurray JJV, Solomon SD; PARAGON-HF Investigators. Health-Related Quality of Life in Heart Failure With Preserved Ejection Fraction: The PARAGON-HF Trial. JACC Heart Fail. 2019 Oct;7(10):862-874. doi: 10.1016/j.jchf.2019.05.015. Epub 2019 Jul 10. PMID 31302043
- [Derived] Balmforth C, Simpson J, Shen L, Jhund PS, Lefkowitz M, Rizkala AR, Rouleau JL, Shi V, Solomon SD, Swedberg K, Zile MR, Packer M, McMurray JJV. Outcomes and Effect of Treatment According to Etiology in HFrEF: An Analysis of PARADIGM-HF. JACC Heart Fail. 2019 Jun;7(6):457-465. doi: 10.1016/j.jchf.2019.02.015. Epub 2019 May 8. PMID 31078482
- [Derived] Myhre PL, Vaduganathan M, Claggett B, Packer M, Desai AS, Rouleau JL, Zile MR, Swedberg K, Lefkowitz M, Shi V, McMurray JJV, Solomon SD. B-Type Natriuretic Peptide During Treatment With Sacubitril/Valsartan: The PARADIGM-HF Trial. J Am Coll Cardiol. 2019 Mar 26;73(11):1264-1272. doi: 10.1016/j.jacc.2019.01.018. Epub 2019 Mar 4. PMID 30846338
- [Derived] Zile MR, O'Meara E, Claggett B, Prescott MF, Solomon SD, Swedberg K, Packer M, McMurray JJV, Shi V, Lefkowitz M, Rouleau J. Effects of Sacubitril/Valsartan on Biomarkers of Extracellular Matrix Regulation in Patients With HFrEF. J Am Coll Cardiol. 2019 Feb 26;73(7):795-806. doi: 10.1016/j.jacc.2018.11.042. PMID 30784673
- [Derived] Bouabdallaoui N, Claggett B, Zile MR, McMurray JJV, O'Meara E, Packer M, Prescott MF, Swedberg K, Solomon SD, Rouleau JL; PARADIGM-HF Investigators and Committees. Growth differentiation factor-15 is not modified by sacubitril/valsartan and is an independent marker of risk in patients with heart failure and reduced ejection fraction: the PARADIGM-HF trial. Eur J Heart Fail. 2018 Dec;20(12):1701-1709. doi: 10.1002/ejhf.1301. Epub 2018 Sep 11. PMID 30204280
- [Derived] O'Meara E, Prescott MF, Claggett B, Rouleau JL, Chiang LM, Solomon SD, Packer M, McMurray JJV, Zile MR. Independent Prognostic Value of Serum Soluble ST2 Measurements in Patients With Heart Failure and a Reduced Ejection Fraction in the PARADIGM-HF Trial (Prospective Comparison of ARNI With ACEI to Determine Impact on Global Mortality and Morbidity in Heart Failure). Circ Heart Fail. 2018 May;11(5):e004446. doi: 10.1161/CIRCHEARTFAILURE.117.004446. PMID 29748349
- [Derived] Packer M, Claggett B, Lefkowitz MP, McMurray JJV, Rouleau JL, Solomon SD, Zile MR. Effect of neprilysin inhibition on renal function in patients with type 2 diabetes and chronic heart failure who are receiving target doses of inhibitors of the renin-angiotensin system: a secondary analysis of the PARADIGM-HF trial. Lancet Diabetes Endocrinol. 2018 Jul;6(7):547-554. doi: 10.1016/S2213-8587(18)30100-1. Epub 2018 Apr 13. PMID 29661699
- [Derived] Chandra A, Lewis EF, Claggett BL, Desai AS, Packer M, Zile MR, Swedberg K, Rouleau JL, Shi VC, Lefkowitz MP, Katova T, McMurray JJV, Solomon SD. Effects of Sacubitril/Valsartan on Physical and Social Activity Limitations in Patients With Heart Failure: A Secondary Analysis of the PARADIGM-HF Trial. JAMA Cardiol. 2018 Jun 1;3(6):498-505. doi: 10.1001/jamacardio.2018.0398. PMID 29617523
- [Derived] Shen L, Ramires F, Martinez F, Bodanese LC, Echeverria LE, Gomez EA, Abraham WT, Dickstein K, Kober L, Packer M, Rouleau JL, Solomon SD, Swedberg K, Zile MR, Jhund PS, Gimpelewicz CR, McMurray JJV; PARADIGM-HF and ATMOSPHERE Investigators and Committees. Contemporary Characteristics and Outcomes in Chagasic Heart Failure Compared With Other Nonischemic and Ischemic Cardiomyopathy. Circ Heart Fail. 2017 Nov;10(11):e004361. doi: 10.1161/CIRCHEARTFAILURE.117.004361. PMID 29141857
- [Derived] Kristensen SL, Jhund PS, Mogensen UM, Rorth R, Abraham WT, Desai A, Dickstein K, Rouleau JL, Zile MR, Swedberg K, Packer M, Solomon SD, Kober L, McMurray JJV; PARADIGM-HF and ATMOSPHERE Committees and Investigators. Prognostic Value of N-Terminal Pro-B-Type Natriuretic Peptide Levels in Heart Failure Patients With and Without Atrial Fibrillation. Circ Heart Fail. 2017 Oct;10(10):e004409. doi: 10.1161/CIRCHEARTFAILURE.117.004409. PMID 29018174
- [Derived] Lewis EF, Claggett BL, McMurray JJV, Packer M, Lefkowitz MP, Rouleau JL, Liu J, Shi VC, Zile MR, Desai AS, Solomon SD, Swedberg K. Health-Related Quality of Life Outcomes in PARADIGM-HF. Circ Heart Fail. 2017 Aug;10(8):e003430. doi: 10.1161/CIRCHEARTFAILURE.116.003430. PMID 28784687
- [Derived] Zile MR, Claggett BL, Prescott MF, McMurray JJ, Packer M, Rouleau JL, Swedberg K, Desai AS, Gong J, Shi VC, Solomon SD. Prognostic Implications of Changes in N-Terminal Pro-B-Type Natriuretic Peptide in Patients With Heart Failure. J Am Coll Cardiol. 2016 Dec 6;68(22):2425-2436. doi: 10.1016/j.jacc.2016.09.931. PMID 27908347
- [Derived] Nadruz W Jr, Claggett BL, McMurray JJ, Packer M, Zile MR, Rouleau JL, Desai AS, Swedberg K, Lefkowitz M, Shi VC, Prescott MF, Solomon SD. Impact of Body Mass Index on the Accuracy of N-Terminal Pro-Brain Natriuretic Peptide and Brain Natriuretic Peptide for Predicting Outcomes in Patients With Chronic Heart Failure and Reduced Ejection Fraction: Insights From the PARADIGM-HF Study (Prospective Comparison of ARNI With ACEI to Determine Impact on Global Mortality and Morbidity in Heart Failure Trial). Circulation. 2016 Nov 29;134(22):1785-1787. doi: 10.1161/CIRCULATIONAHA.116.024976. No abstract available. PMID 27895026
- [Derived] Desai AS, Vardeny O, Claggett B, McMurray JJ, Packer M, Swedberg K, Rouleau JL, Zile MR, Lefkowitz M, Shi V, Solomon SD. Reduced Risk of Hyperkalemia During Treatment of Heart Failure With Mineralocorticoid Receptor Antagonists by Use of Sacubitril/Valsartan Compared With Enalapril: A Secondary Analysis of the PARADIGM-HF Trial. JAMA Cardiol. 2017 Jan 1;2(1):79-85. doi: 10.1001/jamacardio.2016.4733. PMID 27842179
- [Derived] Okumura N, Jhund PS, Gong J, Lefkowitz MP, Rizkala AR, Rouleau JL, Shi VC, Swedberg K, Zile MR, Solomon SD, Packer M, McMurray JJ; PARADIGM-HF Investigators and Committees*. Effects of Sacubitril/Valsartan in the PARADIGM-HF Trial (Prospective Comparison of ARNI with ACEI to Determine Impact on Global Mortality and Morbidity in Heart Failure) According to Background Therapy. Circ Heart Fail. 2016 Sep;9(9):e003212. doi: 10.1161/CIRCHEARTFAILURE.116.003212. PMID 27618854
- [Derived] Solomon SD, Claggett B, Packer M, Desai A, Zile MR, Swedberg K, Rouleau J, Shi V, Lefkowitz M, McMurray JJV. Efficacy of Sacubitril/Valsartan Relative to a Prior Decompensation: The PARADIGM-HF Trial. JACC Heart Fail. 2016 Oct;4(10):816-822. doi: 10.1016/j.jchf.2016.05.002. Epub 2016 Jul 6. PMID 27395349
- [Derived] Kristensen SL, Martinez F, Jhund PS, Arango JL, Belohlavek J, Boytsov S, Cabrera W, Gomez E, Hagege AA, Huang J, Kiatchoosakun S, Kim KS, Mendoza I, Senni M, Squire IB, Vinereanu D, Wong RC, Gong J, Lefkowitz MP, Rizkala AR, Rouleau JL, Shi VC, Solomon SD, Swedberg K, Zile MR, Packer M, McMurray JJ. Geographic variations in the PARADIGM-HF heart failure trial. Eur Heart J. 2016 Nov 1;37(41):3167-3174. doi: 10.1093/eurheartj/ehw226. Epub 2016 Jun 28. PMID 27354044
- [Derived] Desai AS, Solomon S, Claggett B, McMurray JJ, Rouleau J, Swedberg K, Zile M, Lefkowitz M, Shi V, Packer M. Factors Associated With Noncompletion During the Run-In Period Before Randomization and Influence on the Estimated Benefit of LCZ696 in the PARADIGM-HF Trial. Circ Heart Fail. 2016 Jun;9(6):e002735. doi: 10.1161/CIRCHEARTFAILURE.115.002735. PMID 27296397
- [Derived] Okumura N, Jhund PS, Gong J, Lefkowitz MP, Rizkala AR, Rouleau JL, Shi VC, Swedberg K, Zile MR, Solomon SD, Packer M, McMurray JJ; PARADIGM-HF Investigators and Committees*. Importance of Clinical Worsening of Heart Failure Treated in the Outpatient Setting: Evidence From the Prospective Comparison of ARNI With ACEI to Determine Impact on Global Mortality and Morbidity in Heart Failure Trial (PARADIGM-HF). Circulation. 2016 Jun 7;133(23):2254-62. doi: 10.1161/CIRCULATIONAHA.115.020729. Epub 2016 Apr 20. PMID 27143684
- [Derived] Solomon SD, Claggett B, Desai AS, Packer M, Zile M, Swedberg K, Rouleau JL, Shi VC, Starling RC, Kozan O, Dukat A, Lefkowitz MP, McMurray JJ. Influence of Ejection Fraction on Outcomes and Efficacy of Sacubitril/Valsartan (LCZ696) in Heart Failure with Reduced Ejection Fraction: The Prospective Comparison of ARNI with ACEI to Determine Impact on Global Mortality and Morbidity in Heart Failure (PARADIGM-HF) Trial. Circ Heart Fail. 2016 Mar;9(3):e002744. doi: 10.1161/CIRCHEARTFAILURE.115.002744. PMID 26915374
- [Derived] Kristensen SL, Preiss D, Jhund PS, Squire I, Cardoso JS, Merkely B, Martinez F, Starling RC, Desai AS, Lefkowitz MP, Rizkala AR, Rouleau JL, Shi VC, Solomon SD, Swedberg K, Zile MR, McMurray JJ, Packer M; PARADIGM-HF Investigators and Committees. Risk Related to Pre-Diabetes Mellitus and Diabetes Mellitus in Heart Failure With Reduced Ejection Fraction: Insights From Prospective Comparison of ARNI With ACEI to Determine Impact on Global Mortality and Morbidity in Heart Failure Trial. Circ Heart Fail. 2016 Jan;9(1):e002560. doi: 10.1161/CIRCHEARTFAILURE.115.002560. PMID 26754626
- [Derived] Simpson J, Jhund PS, Silva Cardoso J, Martinez F, Mosterd A, Ramires F, Rizkala AR, Senni M, Squire I, Gong J, Lefkowitz MP, Shi VC, Desai AS, Rouleau JL, Swedberg K, Zile MR, McMurray JJV, Packer M, Solomon SD; PARADIGM-HF Investigators and Committees. Comparing LCZ696 with enalapril according to baseline risk using the MAGGIC and EMPHASIS-HF risk scores: an analysis of mortality and morbidity in PARADIGM-HF. J Am Coll Cardiol. 2015 Nov 10;66(19):2059-2071. doi: 10.1016/j.jacc.2015.08.878. PMID 26541915
- [Derived] Andersen MB, Simonsen U, Wehland M, Pietsch J, Grimm D. LCZ696 (Valsartan/Sacubitril)--A Possible New Treatment for Hypertension and Heart Failure. Basic Clin Pharmacol Toxicol. 2016 Jan;118(1):14-22. doi: 10.1111/bcpt.12453. Epub 2015 Sep 4. PMID 26280447
- [Derived] Jhund PS, Fu M, Bayram E, Chen CH, Negrusz-Kawecka M, Rosenthal A, Desai AS, Lefkowitz MP, Rizkala AR, Rouleau JL, Shi VC, Solomon SD, Swedberg K, Zile MR, McMurray JJ, Packer M; PARADIGM-HF Investigators and Committees. Efficacy and safety of LCZ696 (sacubitril-valsartan) according to age: insights from PARADIGM-HF. Eur Heart J. 2015 Oct 7;36(38):2576-84. doi: 10.1093/eurheartj/ehv330. Epub 2015 Jul 31. PMID 26231885
- [Derived] Desai AS, McMurray JJ, Packer M, Swedberg K, Rouleau JL, Chen F, Gong J, Rizkala AR, Brahimi A, Claggett B, Finn PV, Hartley LH, Liu J, Lefkowitz M, Shi V, Zile MR, Solomon SD. Effect of the angiotensin-receptor-neprilysin inhibitor LCZ696 compared with enalapril on mode of death in heart failure patients. Eur Heart J. 2015 Aug 7;36(30):1990-7. doi: 10.1093/eurheartj/ehv186. Epub 2015 May 28. PMID 26022006
- [Derived] McMurray J, Packer M, Desai A, Gong J, Greenlaw N, Lefkowitz M, Rizkala A, Shi V, Rouleau J, Solomon S, Swedberg K, Zile MR, Andersen K, Arango JL, Arnold M, Belohlavek J, Bohm M, Boytsov S, Burgess L, Cabrera W, Chen CH, Erglis A, Fu M, Gomez E, Gonzalez A, Hagege AA, Katova T, Kiatchoosakun S, Kim KS, Bayram E, Martinez F, Merkely B, Mendoza I, Mosterd A, Negrusz-Kawecka M, Peuhkurinen K, Ramires F, Refsgaard J, Senni M, Sibulo AS Jr, Silva-Cardoso J, Squire I, Starling RC, Vinereanu D, Teerlink JR, Wong R; PARADIGM-HF Committees and Investigators. A putative placebo analysis of the effects of LCZ696 on clinical outcomes in heart failure. Eur Heart J. 2015 Feb 14;36(7):434-9. doi: 10.1093/eurheartj/ehu455. PMID 25416329
- [Derived] Packer M, McMurray JJ, Desai AS, Gong J, Lefkowitz MP, Rizkala AR, Rouleau JL, Shi VC, Solomon SD, Swedberg K, Zile M, Andersen K, Arango JL, Arnold JM, Belohlavek J, Bohm M, Boytsov S, Burgess LJ, Cabrera W, Calvo C, Chen CH, Dukat A, Duarte YC, Erglis A, Fu M, Gomez E, Gonzalez-Medina A, Hagege AA, Huang J, Katova T, Kiatchoosakun S, Kim KS, Kozan O, Llamas EB, Martinez F, Merkely B, Mendoza I, Mosterd A, Negrusz-Kawecka M, Peuhkurinen K, Ramires FJ, Refsgaard J, Rosenthal A, Senni M, Sibulo AS Jr, Silva-Cardoso J, Squire IB, Starling RC, Teerlink JR, Vanhaecke J, Vinereanu D, Wong RC; PARADIGM-HF Investigators and Coordinators. Angiotensin receptor neprilysin inhibition compared with enalapril on the risk of clinical progression in surviving patients with heart failure. Circulation. 2015 Jan 6;131(1):54-61. doi: 10.1161/CIRCULATIONAHA.114.013748. Epub 2014 Nov 17. PMID 25403646
- [Derived] McMurray JJ, Packer M, Desai AS, Gong J, Lefkowitz MP, Rizkala AR, Rouleau JL, Shi VC, Solomon SD, Swedberg K, Zile MR; PARADIGM-HF Investigators and Committees. Angiotensin-neprilysin inhibition versus enalapril in heart failure. N Engl J Med. 2014 Sep 11;371(11):993-1004. doi: 10.1056/NEJMoa1409077. Epub 2014 Aug 30. PMID 25176015
- [Derived] McMurray JJ, Packer M, Desai AS, Gong J, Lefkowitz MP, Rizkala AR, Rouleau J, Shi VC, Solomon SD, Swedberg K, Zile MR; PARADIGM-HF Committees and Investigators. Dual angiotensin receptor and neprilysin inhibition as an alternative to angiotensin-converting enzyme inhibition in patients with chronic systolic heart failure: rationale for and design of the Prospective comparison of ARNI with ACEI to Determine Impact on Global Mortality and morbidity in Heart Failure trial (PARADIGM-HF). Eur J Heart Fail. 2013 Sep;15(9):1062-73. doi: 10.1093/eurjhf/hft052. Epub 2013 Apr 5. PMID 23563576

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LCZ696 | Enalapril
Started | 4209 | 4233
GCP Violations | 18 | 19
Mis-randomized | 4 | 2
Full Analysis Set (FAS) | 4187 (patents with GCP violation and mis-randomized are not included in FAS) | 4212 (patents with GCP violation and mis-randomized are not included in FAS)
Completed | 3468 | 3371
Not Completed | 741 | 862
Not completed — Death | 724 | 844
Not completed — Lost to Follow-up | 2 | 5
Not completed — patient's request | 15 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LCZ696 | Enalapril | Total
Number analyzed (Participants) | 4209 | 4233 | 8442
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.78 (11.520) | 63.82 (11.25) | 63.80 (11.385)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 888 | 959 | 1847
  Male | 3321 | 3274 | 6595

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Had First Occurrence of the Composite Endpoint, Which is Defined as Either Cardiovascular (CV) Death or Heart Failure (HF) Hospitalization
Description: Number of participants that had first occurrence of the composite endpoint, which is defined as either CV death or HF hospitalization due to HF.
Time Frame: up to 51 months
Population: Full Analysis Set (FAS) included all randomized patients but the following two exclusions: 6 patients who did not qualify for randomization but were inadvertently randomized into the study and did not receive double-blind study medication; 37 patients because they were randomized at sites that were closed due to serious GCP violations
Measure: Number; unit: participants
Arm/Group | LCZ696 | Enalapril
Number analyzed (Participants) | 4187 | 4212
participants
  Primary Composite | 914 | 1117
  CV death | 558 | 693
  1st HF Hospitalization | 537 | 658

2. Secondary Outcome: Number of Patients - All-cause Mortality
Description: Number of patients - All-cause mortality. All-cause mortality is common in Heart Failure HF patients this measures how many patients had this event. The data is on FAS population up to March 31, 2014
Time Frame: up to 51 months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | LCZ696 | Enalapril
Number analyzed (Participants) | 4187 | 4212
participants | 711 | 835

3. Secondary Outcome: Number of Patients Reported With Adjudicated Primary Causes of Death
Description: Number of patients reported with adjudicated primary causes of death. The data is on Randomization population up to March 31, 2014
Time Frame: up to 51 months
Population: Randomized set (RAN): Consisted of all patients who received a randomization number, regardless of receiving trial medication.
Measure: Number; unit: participants
Arm/Group | LCZ696 | Enalapril
Number analyzed (Participants) | 4209 | 4233
participants
  Number of patients who died | 714 | 837
  CV Death - Fatal MI | 25 | 33
  CV Death - Pump Failure | 147 | 185
  CV Death - Sudden Death | 251 | 311
  CV Death - Presumed Sudden Death | 26 | 23
  CV Death - Presumed CV Death | 67 | 95
  CV Death - Fatal Stroke | 30 | 34
  CV Death - Pulmonary Embolism | 4 | 3
  CV Death - CV procedural | 3 | 4
  Other CV Death | 7 | 6
  Non-CV death - Infection | 36 | 34
  Non-CV death - Malignancy | 41 | 41
  Non-CV death - Renal | 1 | 1
  Non-CV death - Accidental | 13 | 6
  Non-CV death - Pulmonary | 7 | 13
  Non-CV death - Suicide | 4 | 1
  Non-CV death - GI | 16 | 10
  Other Non-CV death | 2 | 4
  Unknown Death | 34 | 33

4. Secondary Outcome: Change From Baseline to Month 8 for the Kansas City Cardiomyopathy Questionnaire (KCCQ) Clinical Summary Score
Description: Change from baseline to Month 8 for the Kansas City Cardiomyopathy Questionnaire (KCCQ) clinical summary score. KCCQ is a 23-item, self-administered instrument that quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life. KCCQ clinical summary score is a composite assessment of physical limitations and total symptom scores. Scores are transformed to a range of 0-100, in which higher scores reflect better health status.
Time Frame: Baseline, Month 8
Population: FAS included all randomized patients with two exclusions: 6 pts who did not qualify for randomization but were misrandomized into the study and did not receive study meds; 37 pts because they were randomized at sites that were closed due to serious GCP violations The analysis included all FAS patients with at least one KCCQ data up-to Month 8.
Measure: Least Squares Mean (Standard Error); unit: KCCQ Score
Arm/Group | LCZ696 | Enalapril
Number analyzed (Participants) | 3833 | 3873
KCCQ Score | -2.99 (0.364) | -4.63 (0.364)

5. Secondary Outcome: Number of Patients With First Confirmed Renal Dysfunction
Description: Number of patients with first confirmed renal dysfunction
Time Frame: up to 51 months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | LCZ696 | Enalapril
Number analyzed (Participants) | 4187 | 4212
participants | 94 | 108

6. Secondary Outcome: Percentage of Participants With New Onset of Atrial Fibrillation (AF)
Description: Percentage of participants with New Onset of Atrial Fibrillation The new onset atrial fibrillation (AF) analysis was based on a subset of FAS: i.e., for patients without a history of AF at baseline (patients with a history of AF were excluded from this analysis).
Time Frame: up to 51 months
Population: The new onset atrial fibrillation (AF) analysis was based on a subset of FAS: i.e., for patients without a history of AF at baseline (patients with a history of AF were excluded from this analysis).
Measure: Number; unit: Percentage of participants
Arm/Group | LCZ696 | Enalapril
Number analyzed (Participants) | 2670 | 2638
Percentage of participants | 3.15 | 3.15

ADVERSE EVENTS:
Description: Safety Population (SAF): Consisted of all randomized patients who received at least one dose of study drug during double-blind period of the study. Patients were analyzed according to the treatment actually received.
Arm/Group | LCZ696 | Enalapril
Serious Adverse Events (participants affected / at risk) | 1937/4203 | 2142/4229
Other Adverse Events (participants affected / at risk) | 2479/4203 | 2594/4229
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LCZ696 (N=4203) | Enalapril (N=4229)
Anaemia (Blood and lymphatic system disorders) | 31 | 47
Anaemia macrocytic (Blood and lymphatic system disorders) | 1 | 0
Anaemia of malignant disease (Blood and lymphatic system disorders) | 1 | 0
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Coagulopathy (Blood and lymphatic system disorders) | 3 | 2
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 2 | 3
Haemorrhagic disorder (Blood and lymphatic system disorders) | 0 | 1
Hypochromic anaemia (Blood and lymphatic system disorders) | 1 | 0
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Microcytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Nephrogenic anaemia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 2 | 2
Pancytopenia (Blood and lymphatic system disorders) | 1 | 1
Pernicious anaemia (Blood and lymphatic system disorders) | 0 | 1
Spontaneous haematoma (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 4
Acute coronary syndrome (Cardiac disorders) | 18 | 18
Acute left ventricular failure (Cardiac disorders) | 4 | 5
Acute myocardial infarction (Cardiac disorders) | 69 | 68
Adams-Stokes syndrome (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 55 | 62
Angina unstable (Cardiac disorders) | 53 | 51
Aortic valve incompetence (Cardiac disorders) | 3 | 4
Aortic valve stenosis (Cardiac disorders) | 0 | 4
Arrhythmia (Cardiac disorders) | 23 | 21
Arrhythmia supraventricular (Cardiac disorders) | 0 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 4 | 4
Arteriospasm coronary (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 108 | 113
Atrial flutter (Cardiac disorders) | 11 | 18
Atrial tachycardia (Cardiac disorders) | 7 | 1
Atrioventricular block (Cardiac disorders) | 2 | 5
Atrioventricular block complete (Cardiac disorders) | 13 | 10
Atrioventricular block first degree (Cardiac disorders) | 1 | 0
Atrioventricular block second degree (Cardiac disorders) | 6 | 5
Atrioventricular dissociation (Cardiac disorders) | 1 | 0
Bradyarrhythmia (Cardiac disorders) | 3 | 4
Bradycardia (Cardiac disorders) | 11 | 13
Bundle branch block left (Cardiac disorders) | 2 | 3
Bundle branch block right (Cardiac disorders) | 0 | 1
Cardiac aneurysm (Cardiac disorders) | 1 | 1
Cardiac arrest (Cardiac disorders) | 30 | 56
Cardiac asthma (Cardiac disorders) | 2 | 3
Cardiac discomfort (Cardiac disorders) | 1 | 3
Cardiac disorder (Cardiac disorders) | 1 | 1
Cardiac failure (Cardiac disorders) | 588 | 649
Cardiac failure acute (Cardiac disorders) | 67 | 93
Cardiac failure chronic (Cardiac disorders) | 112 | 135
Cardiac failure congestive (Cardiac disorders) | 112 | 140
Cardiac fibrillation (Cardiac disorders) | 0 | 1
Cardiac hypertrophy (Cardiac disorders) | 1 | 0
Cardiac perforation (Cardiac disorders) | 1 | 0
Cardiac tamponade (Cardiac disorders) | 0 | 2
Cardiac valve disease (Cardiac disorders) | 0 | 2
Cardiac ventricular thrombosis (Cardiac disorders) | 3 | 3
Cardio-respiratory arrest (Cardiac disorders) | 25 | 27
Cardiogenic shock (Cardiac disorders) | 19 | 38
Cardiomegaly (Cardiac disorders) | 2 | 5
Cardiomyopathy (Cardiac disorders) | 6 | 10
Cardiopulmonary failure (Cardiac disorders) | 7 | 13
Cardiorenal syndrome (Cardiac disorders) | 2 | 2
Cardiovascular disorder (Cardiac disorders) | 1 | 1
Cardiovascular insufficiency (Cardiac disorders) | 1 | 1
Chordae tendinae rupture (Cardiac disorders) | 0 | 1
Congestive cardiomyopathy (Cardiac disorders) | 13 | 29
Cor pulmonale (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 35 | 38
Coronary artery occlusion (Cardiac disorders) | 2 | 1
Coronary artery stenosis (Cardiac disorders) | 5 | 7
Coronary artery thrombosis (Cardiac disorders) | 1 | 1
Defect conduction intraventricular (Cardiac disorders) | 1 | 0
Dilatation atrial (Cardiac disorders) | 0 | 1
Dilatation ventricular (Cardiac disorders) | 1 | 0
Gastrocardiac syndrome (Cardiac disorders) | 0 | 1
Hypertensive cardiomyopathy (Cardiac disorders) | 1 | 0
Hypertensive heart disease (Cardiac disorders) | 1 | 2
Ischaemic cardiomyopathy (Cardiac disorders) | 5 | 14
Left ventricular dysfunction (Cardiac disorders) | 6 | 6
Left ventricular failure (Cardiac disorders) | 9 | 2
Low cardiac output syndrome (Cardiac disorders) | 2 | 2
Mitral valve disease (Cardiac disorders) | 1 | 2
Mitral valve disease mixed (Cardiac disorders) | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 10 | 13
Myocardial infarction (Cardiac disorders) | 65 | 72
Myocardial ischaemia (Cardiac disorders) | 20 | 29
Myocarditis (Cardiac disorders) | 0 | 1
Nodal arrhythmia (Cardiac disorders) | 1 | 1
Nodal rhythm (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 3 | 8
Pericardial effusion (Cardiac disorders) | 1 | 1
Pulseless electrical activity (Cardiac disorders) | 1 | 1
Right ventricular dysfunction (Cardiac disorders) | 1 | 0
Right ventricular failure (Cardiac disorders) | 0 | 4
Sick sinus syndrome (Cardiac disorders) | 10 | 9
Silent myocardial infarction (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 2 | 3
Sinus tachycardia (Cardiac disorders) | 2 | 2
Supraventricular tachycardia (Cardiac disorders) | 9 | 9
Systolic dysfunction (Cardiac disorders) | 0 | 1
Tachyarrhythmia (Cardiac disorders) | 0 | 3
Tachycardia (Cardiac disorders) | 2 | 5
Torsade de pointes (Cardiac disorders) | 0 | 1
Tricuspid valve incompetence (Cardiac disorders) | 0 | 2
Trifascicular block (Cardiac disorders) | 0 | 1
Ventricular arrhythmia (Cardiac disorders) | 5 | 11
Ventricular dysfunction (Cardiac disorders) | 0 | 1
Ventricular dyssynchrony (Cardiac disorders) | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 6 | 4
Ventricular fibrillation (Cardiac disorders) | 22 | 28
Ventricular flutter (Cardiac disorders) | 0 | 1
Ventricular hypokinesia (Cardiac disorders) | 0 | 1
Ventricular tachyarrhythmia (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 66 | 85
Cryptorchism (Congenital, familial and genetic disorders) | 1 | 0
Exomphalos (Congenital, familial and genetic disorders) | 0 | 1
Gastrointestinal arteriovenous malformation (Congenital, familial and genetic disorders) | 0 | 1
Homocystinaemia (Congenital, familial and genetic disorders) | 0 | 1
Hydrocele (Congenital, familial and genetic disorders) | 2 | 0
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 0 | 1
Sickle cell anaemia with crisis (Congenital, familial and genetic disorders) | 0 | 1
Acute vestibular syndrome (Ear and labyrinth disorders) | 1 | 0
Deafness neurosensory (Ear and labyrinth disorders) | 1 | 0
Deafness unilateral (Ear and labyrinth disorders) | 0 | 1
Ear haemorrhage (Ear and labyrinth disorders) | 1 | 0
Mastoid disorder (Ear and labyrinth disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 2 | 0
Vertigo (Ear and labyrinth disorders) | 5 | 9
Vertigo positional (Ear and labyrinth disorders) | 0 | 1
Autoimmune thyroiditis (Endocrine disorders) | 1 | 0
Goitre (Endocrine disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 3 | 3
Hypothyroidism (Endocrine disorders) | 1 | 4
Thyroiditis subacute (Endocrine disorders) | 0 | 1
Amaurosis fugax (Eye disorders) | 1 | 0
Blindness unilateral (Eye disorders) | 0 | 1
Cataract (Eye disorders) | 12 | 8
Cataract diabetic (Eye disorders) | 0 | 1
Conjunctival haemorrhage (Eye disorders) | 0 | 1
Diabetic retinopathy (Eye disorders) | 2 | 1
Diplopia (Eye disorders) | 0 | 1
Glaucoma (Eye disorders) | 1 | 0
Macular oedema (Eye disorders) | 0 | 1
Retinal artery embolism (Eye disorders) | 0 | 1
Retinal detachment (Eye disorders) | 0 | 2
Retinal haemorrhage (Eye disorders) | 1 | 0
Trichiasis (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 2 | 0
Vitreous haemorrhage (Eye disorders) | 0 | 2
Abdominal adhesions (Gastrointestinal disorders) | 1 | 0
Abdominal compartment syndrome (Gastrointestinal disorders) | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 4 | 3
Abdominal hernia (Gastrointestinal disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 15 | 23
Abdominal pain upper (Gastrointestinal disorders) | 6 | 7
Abdominal wall haematoma (Gastrointestinal disorders) | 0 | 1
Acute abdomen (Gastrointestinal disorders) | 1 | 3
Anal fissure (Gastrointestinal disorders) | 2 | 1
Anal fistula (Gastrointestinal disorders) | 2 | 0
Anal haemorrhage (Gastrointestinal disorders) | 0 | 2
Anorectal discomfort (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 5 | 6
Colitis (Gastrointestinal disorders) | 0 | 3
Colitis ischaemic (Gastrointestinal disorders) | 1 | 4
Colitis ulcerative (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 3 | 5
Crohn's disease (Gastrointestinal disorders) | 1 | 0
Dental caries (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 22 | 15
Diverticulum (Gastrointestinal disorders) | 3 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 2
Duodenal stenosis (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 2 | 9
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 3
Duodenal ulcer perforation (Gastrointestinal disorders) | 1 | 0
Duodenitis (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 3 | 4
Dysphagia (Gastrointestinal disorders) | 1 | 1
Enteritis (Gastrointestinal disorders) | 3 | 2
Enterovesical fistula (Gastrointestinal disorders) | 0 | 1
Erosive duodenitis (Gastrointestinal disorders) | 1 | 0
Erosive oesophagitis (Gastrointestinal disorders) | 0 | 3
Faecal incontinence (Gastrointestinal disorders) | 0 | 1
Faecaloma (Gastrointestinal disorders) | 2 | 0
Femoral hernia (Gastrointestinal disorders) | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 3
Gastric hypomotility (Gastrointestinal disorders) | 0 | 1
Gastric perforation (Gastrointestinal disorders) | 1 | 2
Gastric polyps (Gastrointestinal disorders) | 0 | 3
Gastric ulcer (Gastrointestinal disorders) | 3 | 3
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 2
Gastritis (Gastrointestinal disorders) | 7 | 10
Gastritis erosive (Gastrointestinal disorders) | 3 | 4
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 | 1
Gastroduodenal haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastroduodenitis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 22 | 22
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 | 1
Gastrointestinal ulcer (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 | 6
Haematemesis (Gastrointestinal disorders) | 2 | 3
Haematochezia (Gastrointestinal disorders) | 1 | 1
Haemorrhagic erosive gastritis (Gastrointestinal disorders) | 1 | 2
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 2 | 1
Haemorrhoids (Gastrointestinal disorders) | 4 | 2
Hiatus hernia (Gastrointestinal disorders) | 2 | 3
Hyperchlorhydria (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 5 | 2
Ileus paralytic (Gastrointestinal disorders) | 0 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 11 | 17
Inguinal hernia strangulated (Gastrointestinal disorders) | 1 | 2
Inguinal hernia, obstructive (Gastrointestinal disorders) | 2 | 3
Intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 5 | 1
Intestinal obstruction (Gastrointestinal disorders) | 4 | 5
Intestinal perforation (Gastrointestinal disorders) | 1 | 2
Intestinal polyp (Gastrointestinal disorders) | 0 | 1
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 | 1
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 1 | 0
Large intestine polyp (Gastrointestinal disorders) | 5 | 2
Lip oedema (Gastrointestinal disorders) | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 | 2
Melaena (Gastrointestinal disorders) | 3 | 5
Mouth haemorrhage (Gastrointestinal disorders) | 1 | 2
Nausea (Gastrointestinal disorders) | 6 | 6
Obstruction gastric (Gastrointestinal disorders) | 1 | 0
Oesophageal achalasia (Gastrointestinal disorders) | 1 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 0 | 1
Oesophageal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 1 | 1
Pancreatitis (Gastrointestinal disorders) | 2 | 8
Pancreatitis acute (Gastrointestinal disorders) | 7 | 4
Pancreatitis chronic (Gastrointestinal disorders) | 1 | 0
Parotid duct obstruction (Gastrointestinal disorders) | 0 | 2
Parotid gland enlargement (Gastrointestinal disorders) | 0 | 1
Peptic ulcer (Gastrointestinal disorders) | 2 | 1
Peptic ulcer perforation (Gastrointestinal disorders) | 1 | 0
Portal hypertensive gastropathy (Gastrointestinal disorders) | 0 | 2
Proctalgia (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 8 | 3
Rectal polyp (Gastrointestinal disorders) | 2 | 1
Rectal prolapse (Gastrointestinal disorders) | 1 | 0
Rectal stenosis (Gastrointestinal disorders) | 0 | 1
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 | 0
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 3 | 3
Stomatitis (Gastrointestinal disorders) | 0 | 1
Subileus (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 2 | 1
Umbilical hernia (Gastrointestinal disorders) | 0 | 6
Umbilical hernia, obstructive (Gastrointestinal disorders) | 2 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 9 | 6
Varices oesophageal (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 10 | 14
Accidental death (General disorders) | 2 | 0
Asthenia (General disorders) | 9 | 9
Cardiac complication associated with device (General disorders) | 1 | 1
Cardiac death (General disorders) | 85 | 114
Chest discomfort (General disorders) | 3 | 1
Chest pain (General disorders) | 3 | 3
Chills (General disorders) | 0 | 1
Concomitant disease aggravated (General disorders) | 1 | 0
Death (General disorders) | 56 | 78
Device battery issue (General disorders) | 11 | 8
Device breakage (General disorders) | 1 | 0
Device dislocation (General disorders) | 3 | 3
Device failure (General disorders) | 6 | 5
Device issue (General disorders) | 1 | 2
Device lead damage (General disorders) | 2 | 1
Device leakage (General disorders) | 0 | 1
Device malfunction (General disorders) | 15 | 11
Device occlusion (General disorders) | 1 | 2
Device stimulation issue (General disorders) | 0 | 1
Disease progression (General disorders) | 1 | 0
Drowning (General disorders) | 0 | 1
Euthanasia (General disorders) | 1 | 0
Exercise tolerance decreased (General disorders) | 1 | 1
Fatigue (General disorders) | 1 | 10
Gait disturbance (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 2 | 3
Generalised oedema (General disorders) | 0 | 1
Hernia (General disorders) | 1 | 1
Hernia obstructive (General disorders) | 0 | 1
Hyperthermia (General disorders) | 1 | 0
Impaired healing (General disorders) | 1 | 1
Implant site haematoma (General disorders) | 0 | 1
Implant site inflammation (General disorders) | 1 | 0
Implant site reaction (General disorders) | 1 | 0
Implant site ulcer (General disorders) | 1 | 1
Inflammation (General disorders) | 1 | 0
Local swelling (General disorders) | 0 | 3
Malaise (General disorders) | 4 | 2
Medical device complication (General disorders) | 5 | 1
Medical device pain (General disorders) | 0 | 3
Medical device site reaction (General disorders) | 0 | 1
Multi-organ disorder (General disorders) | 1 | 0
Multi-organ failure (General disorders) | 14 | 15
Necrosis (General disorders) | 1 | 1
Non-cardiac chest pain (General disorders) | 33 | 36
Oedema (General disorders) | 0 | 1
Oedema due to cardiac disease (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 10 | 15
Pacemaker generated arrhythmia (General disorders) | 0 | 1
Perforated ulcer (General disorders) | 0 | 1
Pyrexia (General disorders) | 9 | 12
Sudden cardiac death (General disorders) | 67 | 69
Sudden death (General disorders) | 66 | 78
Temperature regulation disorder (General disorders) | 0 | 1
Vessel puncture site haematoma (General disorders) | 1 | 0
Vessel puncture site haemorrhage (General disorders) | 0 | 1
Acute hepatic failure (Hepatobiliary disorders) | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 4 | 3
Biliary colic (Hepatobiliary disorders) | 0 | 2
Biliary dilatation (Hepatobiliary disorders) | 2 | 0
Cardiac cirrhosis (Hepatobiliary disorders) | 1 | 1
Cholangitis (Hepatobiliary disorders) | 2 | 1
Cholangitis acute (Hepatobiliary disorders) | 4 | 0
Cholecystitis (Hepatobiliary disorders) | 5 | 8
Cholecystitis acute (Hepatobiliary disorders) | 12 | 12
Cholecystitis chronic (Hepatobiliary disorders) | 3 | 1
Cholelithiasis (Hepatobiliary disorders) | 10 | 17
Cholestasis (Hepatobiliary disorders) | 0 | 2
Gallbladder perforation (Hepatobiliary disorders) | 0 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 3 | 5
Hepatic congestion (Hepatobiliary disorders) | 0 | 3
Hepatic failure (Hepatobiliary disorders) | 5 | 4
Hepatic function abnormal (Hepatobiliary disorders) | 3 | 2
Hepatic ischaemia (Hepatobiliary disorders) | 1 | 0
Hepatic steatosis (Hepatobiliary disorders) | 3 | 1
Hepatitis (Hepatobiliary disorders) | 2 | 1
Hepatitis acute (Hepatobiliary disorders) | 1 | 0
Hepatitis toxic (Hepatobiliary disorders) | 0 | 1
Hepatocellular injury (Hepatobiliary disorders) | 0 | 1
Hepatomegaly (Hepatobiliary disorders) | 0 | 2
Hepatorenal syndrome (Hepatobiliary disorders) | 0 | 1
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0
Hydrocholecystis (Hepatobiliary disorders) | 1 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 2
Ischaemic hepatitis (Hepatobiliary disorders) | 0 | 2
Jaundice (Hepatobiliary disorders) | 5 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 1
Liver disorder (Hepatobiliary disorders) | 0 | 2
Liver injury (Hepatobiliary disorders) | 1 | 2
Portal hypertension (Hepatobiliary disorders) | 0 | 1
Portal vein thrombosis (Hepatobiliary disorders) | 1 | 0
Allergy to arthropod sting (Immune system disorders) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 2 | 0
Anaphylactic shock (Immune system disorders) | 1 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 5
Hypersensitivity (Immune system disorders) | 2 | 0
Sarcoidosis (Immune system disorders) | 2 | 0
Abdominal abscess (Infections and infestations) | 0 | 1
Abdominal wall abscess (Infections and infestations) | 0 | 1
Abdominal wall infection (Infections and infestations) | 1 | 0
Abscess limb (Infections and infestations) | 1 | 1
Abscess neck (Infections and infestations) | 1 | 2
Abscess oral (Infections and infestations) | 0 | 1
Acinetobacter bacteraemia (Infections and infestations) | 0 | 1
Acinetobacter infection (Infections and infestations) | 0 | 1
Acute endocarditis (Infections and infestations) | 2 | 2
Acute tonsillitis (Infections and infestations) | 0 | 1
American trypanosomiasis (Infections and infestations) | 0 | 1
Anal abscess (Infections and infestations) | 1 | 3
Appendicitis (Infections and infestations) | 5 | 6
Appendicitis perforated (Infections and infestations) | 2 | 1
Arthritis bacterial (Infections and infestations) | 1 | 0
Arthritis infective (Infections and infestations) | 1 | 2
Atypical pneumonia (Infections and infestations) | 2 | 1
Bacteraemia (Infections and infestations) | 2 | 0
Bacterial diarrhoea (Infections and infestations) | 0 | 1
Bacterial infection (Infections and infestations) | 0 | 1
Bacterial prostatitis (Infections and infestations) | 0 | 1
Bacterial sepsis (Infections and infestations) | 0 | 1
Bacterial tracheitis (Infections and infestations) | 0 | 1
Bacteriuria (Infections and infestations) | 0 | 1
Biliary sepsis (Infections and infestations) | 2 | 1
Breast cellulitis (Infections and infestations) | 1 | 0
Bronchiolitis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 20 | 26
Bronchitis bacterial (Infections and infestations) | 1 | 1
Bronchitis fungal (Infections and infestations) | 1 | 0
Bronchitis viral (Infections and infestations) | 1 | 1
Bronchopneumonia (Infections and infestations) | 21 | 14
Campylobacter gastroenteritis (Infections and infestations) | 1 | 1
Carbuncle (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 19 | 23
Cellulitis staphylococcal (Infections and infestations) | 0 | 1
Cholecystitis infective (Infections and infestations) | 2 | 0
Chronic hepatitis B (Infections and infestations) | 0 | 1
Clostridial infection (Infections and infestations) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 3 | 2
Clostridium difficile infection (Infections and infestations) | 0 | 3
Cystitis (Infections and infestations) | 1 | 5
Cytomegalovirus infection (Infections and infestations) | 0 | 1
Dacryocanaliculitis (Infections and infestations) | 0 | 1
Dermatophytosis (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 10 | 11
Device related sepsis (Infections and infestations) | 0 | 1
Diabetic foot infection (Infections and infestations) | 2 | 1
Diabetic gangrene (Infections and infestations) | 2 | 0
Diarrhoea infectious (Infections and infestations) | 1 | 1
Disseminated tuberculosis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 2 | 3
Empyema (Infections and infestations) | 0 | 1
Encephalitis (Infections and infestations) | 0 | 1
Encephalitis viral (Infections and infestations) | 1 | 0
Endocarditis (Infections and infestations) | 4 | 8
Endocarditis bacterial (Infections and infestations) | 1 | 0
Epididymitis (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 10 | 11
Escherichia sepsis (Infections and infestations) | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 2
Gallbladder abscess (Infections and infestations) | 0 | 1
Gangrene (Infections and infestations) | 8 | 12
Gastroenteritis (Infections and infestations) | 22 | 22
Gastroenteritis clostridial (Infections and infestations) | 2 | 0
Gastroenteritis norovirus (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 1
Gastrointestinal bacterial infection (Infections and infestations) | 0 | 1
Gastrointestinal infection (Infections and infestations) | 1 | 2
Gastrointestinal viral infection (Infections and infestations) | 1 | 0
Groin abscess (Infections and infestations) | 2 | 0
H1N1 influenza (Infections and infestations) | 0 | 2
Haematoma infection (Infections and infestations) | 1 | 0
Haemorrhagic fever (Infections and infestations) | 1 | 0
Hepatitis A (Infections and infestations) | 0 | 2
Hepatitis B (Infections and infestations) | 1 | 1
Herpes simplex meningoencephalitis (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 3
Implant site infection (Infections and infestations) | 3 | 1
Infected cyst (Infections and infestations) | 0 | 1
Infected dermal cyst (Infections and infestations) | 1 | 0
Infected skin ulcer (Infections and infestations) | 1 | 3
Infectious pleural effusion (Infections and infestations) | 1 | 1
Infective exacerbation of bronchiectasis (Infections and infestations) | 0 | 2
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 5 | 3
Influenza (Infections and infestations) | 5 | 5
Intervertebral discitis (Infections and infestations) | 2 | 0
Joint abscess (Infections and infestations) | 0 | 1
Kidney infection (Infections and infestations) | 0 | 1
Labyrinthitis (Infections and infestations) | 0 | 1
Laryngitis (Infections and infestations) | 0 | 1
Liver abscess (Infections and infestations) | 1 | 0
Lobar pneumonia (Infections and infestations) | 5 | 6
Localised infection (Infections and infestations) | 4 | 2
Lower respiratory tract infection (Infections and infestations) | 13 | 21
Lower respiratory tract infection bacterial (Infections and infestations) | 0 | 1
Lower respiratory tract infection viral (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 6 | 12
Meningitis (Infections and infestations) | 0 | 1
Morganella infection (Infections and infestations) | 0 | 1
Myocarditis infectious (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 2
Necrotising fasciitis (Infections and infestations) | 3 | 0
Orchitis (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 7 | 2
Otitis media (Infections and infestations) | 0 | 1
Parotitis (Infections and infestations) | 0 | 1
Perineal abscess (Infections and infestations) | 1 | 0
Peritoneal abscess (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 6 | 2
Pharyngitis (Infections and infestations) | 0 | 1
Pneumococcal sepsis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 155 | 181
Pneumonia bacterial (Infections and infestations) | 3 | 1
Pneumonia haemophilus (Infections and infestations) | 1 | 0
Pneumonia influenzal (Infections and infestations) | 0 | 1
Pneumonia klebsiella (Infections and infestations) | 0 | 1
Pneumonia legionella (Infections and infestations) | 0 | 1
Pneumonia pneumococcal (Infections and infestations) | 0 | 1
Pneumonia staphylococcal (Infections and infestations) | 1 | 0
Pneumonia viral (Infections and infestations) | 1 | 0
Post procedural infection (Infections and infestations) | 2 | 0
Post procedural pneumonia (Infections and infestations) | 0 | 1
Postoperative wound infection (Infections and infestations) | 1 | 3
Pseudomembranous colitis (Infections and infestations) | 1 | 0
Pulmonary sepsis (Infections and infestations) | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 5 | 2
Pyelonephritis (Infections and infestations) | 3 | 2
Pyelonephritis acute (Infections and infestations) | 1 | 3
Pyelonephritis chronic (Infections and infestations) | 2 | 1
Rabies (Infections and infestations) | 1 | 0
Rectal abscess (Infections and infestations) | 1 | 2
Respiratory syncytial virus infection (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 15 | 8
Respiratory tract infection bacterial (Infections and infestations) | 0 | 1
Salmonellosis (Infections and infestations) | 1 | 0
Scrotal gangrene (Infections and infestations) | 0 | 1
Scrotal infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 24 | 37
Septic shock (Infections and infestations) | 17 | 23
Sinusitis (Infections and infestations) | 0 | 1
Skin bacterial infection (Infections and infestations) | 1 | 0
Soft tissue infection (Infections and infestations) | 0 | 2
Staphylococcal abscess (Infections and infestations) | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 1 | 2
Staphylococcal infection (Infections and infestations) | 0 | 4
Staphylococcal sepsis (Infections and infestations) | 4 | 0
Stoma site infection (Infections and infestations) | 0 | 1
Streptococcal bacteraemia (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 2
Tooth abscess (Infections and infestations) | 1 | 1
Tooth infection (Infections and infestations) | 0 | 1
Tracheobronchitis (Infections and infestations) | 2 | 3
Tuberculosis (Infections and infestations) | 0 | 1
Tuberculous pleurisy (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 6 | 11
Urinary tract infection (Infections and infestations) | 41 | 34
Urinary tract infection bacterial (Infections and infestations) | 2 | 2
Urosepsis (Infections and infestations) | 8 | 9
Vestibular neuronitis (Infections and infestations) | 1 | 1
Viraemia (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 1 | 4
Viral myocarditis (Infections and infestations) | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 2
Wound abscess (Infections and infestations) | 1 | 1
Wound sepsis (Infections and infestations) | 1 | 0
Abdominal injury (Injury, poisoning and procedural complications) | 1 | 1
Accident (Injury, poisoning and procedural complications) | 0 | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 | 2
Animal bite (Injury, poisoning and procedural complications) | 1 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 2
Arterial restenosis (Injury, poisoning and procedural complications) | 0 | 1
Bone contusion (Injury, poisoning and procedural complications) | 0 | 1
Brain contusion (Injury, poisoning and procedural complications) | 1 | 2
Cardiac contusion (Injury, poisoning and procedural complications) | 0 | 1
Cardiac function disturbance postoperative (Injury, poisoning and procedural complications) | 0 | 3
Cardiac valve replacement complication (Injury, poisoning and procedural complications) | 0 | 1
Cardiac valve rupture (Injury, poisoning and procedural complications) | 1 | 1
Chemical peritonitis (Injury, poisoning and procedural complications) | 1 | 1
Chest injury (Injury, poisoning and procedural complications) | 2 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 2 | 1
Compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 4
Coronary artery restenosis (Injury, poisoning and procedural complications) | 1 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 1
Cystitis radiation (Injury, poisoning and procedural complications) | 1 | 0
Excoriation (Injury, poisoning and procedural complications) | 1 | 1
Extradural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Eyeball rupture (Injury, poisoning and procedural complications) | 0 | 1
Face injury (Injury, poisoning and procedural complications) | 0 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 2 | 1
Fall (Injury, poisoning and procedural complications) | 6 | 10
Femoral neck fracture (Injury, poisoning and procedural complications) | 5 | 7
Femur fracture (Injury, poisoning and procedural complications) | 6 | 7
Fibula fracture (Injury, poisoning and procedural complications) | 2 | 2
Foot fracture (Injury, poisoning and procedural complications) | 0 | 2
Forearm fracture (Injury, poisoning and procedural complications) | 1 | 0
Foreign body (Injury, poisoning and procedural complications) | 1 | 0
Graft complication (Injury, poisoning and procedural complications) | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 1 | 1
Head injury (Injury, poisoning and procedural complications) | 6 | 5
Hip fracture (Injury, poisoning and procedural complications) | 6 | 12
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 3
Incisional hernia (Injury, poisoning and procedural complications) | 3 | 1
Jaw fracture (Injury, poisoning and procedural complications) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 4 | 0
Laceration (Injury, poisoning and procedural complications) | 5 | 1
Limb traumatic amputation (Injury, poisoning and procedural complications) | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 2 | 2
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 2 | 1
Median nerve injury (Injury, poisoning and procedural complications) | 1 | 0
Medication error (Injury, poisoning and procedural complications) | 0 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 2
Multiple fractures (Injury, poisoning and procedural complications) | 1 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 1 | 1
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 3 | 5
Patella fracture (Injury, poisoning and procedural complications) | 1 | 3
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0
Post concussion syndrome (Injury, poisoning and procedural complications) | 1 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 2 | 2
Post procedural discharge (Injury, poisoning and procedural complications) | 0 | 1
Post procedural fistula (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 2
Post procedural myocardial infarction (Injury, poisoning and procedural complications) | 1 | 1
Postoperative renal failure (Injury, poisoning and procedural complications) | 1 | 0
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 1 | 0
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 | 0
Procedural complication (Injury, poisoning and procedural complications) | 0 | 1
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Pubis fracture (Injury, poisoning and procedural complications) | 1 | 1
Radiation proctitis (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 4 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 7 | 3
Sacroiliac fracture (Injury, poisoning and procedural complications) | 1 | 0
Scapula fracture (Injury, poisoning and procedural complications) | 0 | 1
Seroma (Injury, poisoning and procedural complications) | 1 | 0
Skull fracture (Injury, poisoning and procedural complications) | 0 | 2
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 3 | 4
Spinal cord injury lumbar (Injury, poisoning and procedural complications) | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 2 | 3
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 11 | 5
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 2
Tendon rupture (Injury, poisoning and procedural complications) | 3 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 3
Tibia fracture (Injury, poisoning and procedural complications) | 2 | 2
Toxicity to various agents (Injury, poisoning and procedural complications) | 8 | 9
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 2
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Vascular graft complication (Injury, poisoning and procedural complications) | 2 | 0
Vascular graft occlusion (Injury, poisoning and procedural complications) | 2 | 0
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 1 | 0
Vascular procedure complication (Injury, poisoning and procedural complications) | 1 | 0
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Wound necrosis (Injury, poisoning and procedural complications) | 1 | 1
Acid base balance abnormal (Investigations) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood albumin decreased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 4 | 2
Blood glucose increased (Investigations) | 2 | 0
Blood potassium decreased (Investigations) | 0 | 1
Blood pressure decreased (Investigations) | 1 | 0
Blood pressure systolic decreased (Investigations) | 0 | 1
Blood sodium decreased (Investigations) | 1 | 0
C-reactive protein increased (Investigations) | 0 | 1
Cardiac function test abnormal (Investigations) | 0 | 1
Coagulation factor increased (Investigations) | 0 | 1
Coagulation time prolonged (Investigations) | 1 | 0
Creatinine renal clearance decreased (Investigations) | 0 | 1
Ejection fraction (Investigations) | 1 | 0
Ejection fraction decreased (Investigations) | 2 | 2
Electrocardiogram QRS complex abnormal (Investigations) | 0 | 1
Escherichia test positive (Investigations) | 0 | 1
Gastric pH decreased (Investigations) | 0 | 2
Glomerular filtration rate decreased (Investigations) | 2 | 1
Haemoglobin decreased (Investigations) | 1 | 2
Heart rate decreased (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 2 | 0
International normalised ratio abnormal (Investigations) | 0 | 2
International normalised ratio increased (Investigations) | 1 | 8
Liver function test abnormal (Investigations) | 1 | 3
Oxygen saturation decreased (Investigations) | 1 | 0
Prothrombin time abnormal (Investigations) | 1 | 0
Prothrombin time prolonged (Investigations) | 0 | 1
Respiratory rate increased (Investigations) | 1 | 0
Troponin increased (Investigations) | 0 | 1
Urine output decreased (Investigations) | 1 | 0
Venous pressure jugular increased (Investigations) | 0 | 1
Weight decreased (Investigations) | 5 | 5
Weight increased (Investigations) | 1 | 2
Cachexia (Metabolism and nutrition disorders) | 3 | 1
Decreased appetite (Metabolism and nutrition disorders) | 4 | 5
Dehydration (Metabolism and nutrition disorders) | 22 | 29
Diabetes mellitus (Metabolism and nutrition disorders) | 24 | 23
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 7 | 8
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 4
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 2
Failure to thrive (Metabolism and nutrition disorders) | 2 | 0
Fluid overload (Metabolism and nutrition disorders) | 2 | 2
Gout (Metabolism and nutrition disorders) | 7 | 10
Hyperglycaemia (Metabolism and nutrition disorders) | 6 | 4
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 17 | 42
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 2
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 1
Hypochloraemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 15 | 14
Hypokalaemia (Metabolism and nutrition disorders) | 12 | 9
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 6 | 12
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 3 | 2
Insulin resistance (Metabolism and nutrition disorders) | 1 | 0
Iron deficiency (Metabolism and nutrition disorders) | 1 | 1
Iron overload (Metabolism and nutrition disorders) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 2 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 3
Metabolic disorder (Metabolism and nutrition disorders) | 1 | 1
Mineral deficiency (Metabolism and nutrition disorders) | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 2 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 1
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1 | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 3 | 2
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 1
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 | 2
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc displacement (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 | 2
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint laxity (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 3 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 3 | 1
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle necrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle swelling (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 4
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 4 | 5
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Myalgia intercostal (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 16 | 15
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 | 2
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 2
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 3
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 4 | 2
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 3
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 3
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 | 1
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 8
Adenosquamous cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 7
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign neoplasm of adrenal gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Benign salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Biliary neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder adenocarcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 | 5
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Bone cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 3
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 4
Bronchioloalveolar carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Chronic myelomonocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 11
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Gastrointestinal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hypergammaglobulinaemia benign monoclonal (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hypopharyngeal neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Inflammatory carcinoma of the breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Large intestine benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Laryngeal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Laryngeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Liposarcoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 | 13
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant mediastinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Malignant neoplasm of pleura (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 6
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 1
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Metastases to spleen (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Nasal neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Nasopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neurilemmoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 2
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 14
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 6
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Refractory cytopenia with unilineage dysplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 4
Renal cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Salivary gland adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Soft tissue cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Spermatocytic seminoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 3
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Tumour ulceration (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Amnesia (Nervous system disorders) | 0 | 1
Aphasia (Nervous system disorders) | 2 | 0
Ataxia (Nervous system disorders) | 1 | 0
Basilar artery thrombosis (Nervous system disorders) | 0 | 1
Brain hypoxia (Nervous system disorders) | 1 | 1
Brain injury (Nervous system disorders) | 2 | 1
Brain mass (Nervous system disorders) | 0 | 1
Brain oedema (Nervous system disorders) | 1 | 4
Brain stem infarction (Nervous system disorders) | 1 | 1
Carotid artery disease (Nervous system disorders) | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 4 | 2
Carpal tunnel syndrome (Nervous system disorders) | 1 | 1
Cerebellar atrophy (Nervous system disorders) | 1 | 0
Cerebellar infarction (Nervous system disorders) | 2 | 1
Cerebral atrophy (Nervous system disorders) | 1 | 0
Cerebral haematoma (Nervous system disorders) | 0 | 3
Cerebral haemorrhage (Nervous system disorders) | 5 | 6
Cerebral infarction (Nervous system disorders) | 8 | 13
Cerebral ischaemia (Nervous system disorders) | 1 | 2
Cerebral venous thrombosis (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 71 | 72
Cerebrovascular disorder (Nervous system disorders) | 1 | 1
Cerebrovascular insufficiency (Nervous system disorders) | 2 | 1
Coma (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 5 | 7
Convulsions local (Nervous system disorders) | 1 | 0
Dementia (Nervous system disorders) | 2 | 2
Dementia Alzheimer's type (Nervous system disorders) | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 2
Diabetic coma (Nervous system disorders) | 2 | 0
Diabetic neuropathy (Nervous system disorders) | 2 | 2
Dizziness (Nervous system disorders) | 10 | 5
Dysarthria (Nervous system disorders) | 2 | 3
Embolic stroke (Nervous system disorders) | 3 | 6
Encephalomalacia (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 3 | 1
Guillain-Barre syndrome (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 4 | 0
Haemorrhagic stroke (Nervous system disorders) | 5 | 5
Haemorrhagic transformation stroke (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 3 | 0
Hemiparesis (Nervous system disorders) | 3 | 1
Hemiplegia (Nervous system disorders) | 1 | 3
Hemisensory neglect (Nervous system disorders) | 0 | 1
Hepatic encephalopathy (Nervous system disorders) | 0 | 1
Hydrocephalus (Nervous system disorders) | 1 | 0
Hyperaesthesia (Nervous system disorders) | 0 | 1
Hypercapnic coma (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 2
Hypoglycaemic coma (Nervous system disorders) | 1 | 1
Hypoglycaemic seizure (Nervous system disorders) | 0 | 1
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 | 2
Intercostal neuralgia (Nervous system disorders) | 0 | 1
Ischaemic neuropathy (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 40 | 37
Lacunar infarction (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 2 | 4
Mental retardation (Nervous system disorders) | 1 | 0
Metabolic encephalopathy (Nervous system disorders) | 0 | 1
Motor dysfunction (Nervous system disorders) | 1 | 0
Movement disorder (Nervous system disorders) | 0 | 1
Multiple system atrophy (Nervous system disorders) | 1 | 0
Neuralgia (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 3
Paraparesis (Nervous system disorders) | 0 | 1
Parkinson's disease (Nervous system disorders) | 1 | 0
Partial seizures (Nervous system disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1
Polyneuropathy (Nervous system disorders) | 1 | 0
Presenile dementia (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 5 | 7
Radiculopathy (Nervous system disorders) | 2 | 0
Reversible ischaemic neurological deficit (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 1 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 3 | 5
Syncope (Nervous system disorders) | 43 | 68
Tension headache (Nervous system disorders) | 1 | 0
Toxic encephalopathy (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 18 | 22
VIIth nerve paralysis (Nervous system disorders) | 0 | 2
Vertebral artery stenosis (Nervous system disorders) | 1 | 0
Vertebrobasilar insufficiency (Nervous system disorders) | 4 | 1
Vocal cord paralysis (Nervous system disorders) | 0 | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 2 | 0
Alcohol abuse (Psychiatric disorders) | 0 | 1
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 | 0
Alcoholism (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 3 | 2
Completed suicide (Psychiatric disorders) | 2 | 1
Confusional state (Psychiatric disorders) | 6 | 8
Delirium (Psychiatric disorders) | 2 | 4
Delirium tremens (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 5 | 0
Disorientation (Psychiatric disorders) | 0 | 2
Emotional distress (Psychiatric disorders) | 0 | 1
Generalised anxiety disorder (Psychiatric disorders) | 1 | 0
Hallucination (Psychiatric disorders) | 0 | 2
Hypochondriasis (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 2
Major depression (Psychiatric disorders) | 0 | 1
Mental disorder (Psychiatric disorders) | 2 | 1
Mental disorder due to a general medical condition (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 4 | 0
Mood disorder due to a general medical condition (Psychiatric disorders) | 0 | 1
Panic disorder (Psychiatric disorders) | 1 | 1
Psychiatric symptom (Psychiatric disorders) | 0 | 1
Psychotic disorder (Psychiatric disorders) | 0 | 2
Psychotic disorder due to a general medical condition (Psychiatric disorders) | 0 | 1
Schizophrenia (Psychiatric disorders) | 0 | 1
Somatisation disorder (Psychiatric disorders) | 1 | 0
Somatoform disorder cardiovascular (Psychiatric disorders) | 0 | 1
Somatoform disorder gastrointestinal (Psychiatric disorders) | 0 | 1
Suicide attempt (Psychiatric disorders) | 1 | 1
Acute prerenal failure (Renal and urinary disorders) | 0 | 1
Azotaemia (Renal and urinary disorders) | 1 | 0
Bladder diverticulum (Renal and urinary disorders) | 1 | 0
Calculus ureteric (Renal and urinary disorders) | 2 | 0
Crush syndrome (Renal and urinary disorders) | 1 | 0
Cystitis erosive (Renal and urinary disorders) | 0 | 1
Cystitis haemorrhagic (Renal and urinary disorders) | 1 | 0
Cystitis noninfective (Renal and urinary disorders) | 0 | 2
Diabetic nephropathy (Renal and urinary disorders) | 0 | 2
Dysuria (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 14 | 10
Hydronephrosis (Renal and urinary disorders) | 0 | 3
Incontinence (Renal and urinary disorders) | 0 | 1
Kidney fibrosis (Renal and urinary disorders) | 0 | 1
Lower urinary tract symptoms (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 2 | 4
Nephropathy (Renal and urinary disorders) | 1 | 0
Nephropathy toxic (Renal and urinary disorders) | 0 | 1
Nephrosclerosis (Renal and urinary disorders) | 2 | 0
Nephrotic syndrome (Renal and urinary disorders) | 1 | 2
Oliguria (Renal and urinary disorders) | 0 | 1
Pelvi-ureteric obstruction (Renal and urinary disorders) | 1 | 0
Prerenal failure (Renal and urinary disorders) | 1 | 3
Proteinuria (Renal and urinary disorders) | 2 | 0
Renal aneurysm (Renal and urinary disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 2 | 1
Renal cyst (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 43 | 54
Renal failure acute (Renal and urinary disorders) | 74 | 79
Renal failure chronic (Renal and urinary disorders) | 9 | 13
Renal impairment (Renal and urinary disorders) | 46 | 57
Renal injury (Renal and urinary disorders) | 2 | 0
Renal tubular acidosis (Renal and urinary disorders) | 0 | 1
Renal tubular necrosis (Renal and urinary disorders) | 1 | 1
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 | 3
Urethral stenosis (Renal and urinary disorders) | 2 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 2
Urinary retention (Renal and urinary disorders) | 10 | 8
Urine flow decreased (Renal and urinary disorders) | 0 | 1
Acquired phimosis (Reproductive system and breast disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 8 | 9
Breast pain (Reproductive system and breast disorders) | 1 | 0
Cervical polyp (Reproductive system and breast disorders) | 1 | 1
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1
Perineal pain (Reproductive system and breast disorders) | 1 | 1
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Prostatic obstruction (Reproductive system and breast disorders) | 1 | 1
Prostatitis (Reproductive system and breast disorders) | 3 | 3
Uterine haemorrhage (Reproductive system and breast disorders) | 1 | 0
Uterine polyp (Reproductive system and breast disorders) | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1
Vaginal relaxation (Reproductive system and breast disorders) | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 20 | 19
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 11 | 11
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 | 6
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 3 | 6
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 40 | 46
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 9
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 51 | 57
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Dyspnoea paroxysmal nocturnal (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 | 7
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 | 11
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 7
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nocturnal dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 16 | 19
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 5 | 8
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 6 | 3
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 6
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 22 | 23
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary microemboli (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 21 | 21
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 25 | 26
Respiratory fatigue (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Vocal cord leukoplakia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 3 | 4
Angiokeratoma (Skin and subcutaneous tissue disorders) | 0 | 1
Cutaneous vasculitis (Skin and subcutaneous tissue disorders) | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 2 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 7 | 7
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 2
Hypersensitivity vasculitis (Skin and subcutaneous tissue disorders) | 0 | 1
Lichen planus (Skin and subcutaneous tissue disorders) | 0 | 1
Pemphigoid (Skin and subcutaneous tissue disorders) | 1 | 0
Pemphigus (Skin and subcutaneous tissue disorders) | 0 | 1
Penile ulceration (Skin and subcutaneous tissue disorders) | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Skin burning sensation (Skin and subcutaneous tissue disorders) | 1 | 0
Skin erosion (Skin and subcutaneous tissue disorders) | 0 | 1
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 3 | 6
Skin ulcer haemorrhage (Skin and subcutaneous tissue disorders) | 1 | 0
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Cardiac pacemaker insertion (Surgical and medical procedures) | 0 | 1
Endotracheal intubation (Surgical and medical procedures) | 0 | 1
Implantable defibrillator insertion (Surgical and medical procedures) | 1 | 0
Lymphadenectomy (Surgical and medical procedures) | 0 | 1
Resuscitation (Surgical and medical procedures) | 1 | 1
Thyroidectomy (Surgical and medical procedures) | 0 | 1
Accelerated hypertension (Vascular disorders) | 0 | 2
Aneurysm (Vascular disorders) | 0 | 1
Angiodysplasia (Vascular disorders) | 0 | 1
Aortic aneurysm (Vascular disorders) | 8 | 11
Aortic dilatation (Vascular disorders) | 1 | 0
Aortic occlusion (Vascular disorders) | 1 | 0
Aortic stenosis (Vascular disorders) | 6 | 2
Arterial occlusive disease (Vascular disorders) | 1 | 0
Arterial thrombosis (Vascular disorders) | 0 | 1
Arteriosclerosis (Vascular disorders) | 3 | 1
Arteriovenous fistula (Vascular disorders) | 1 | 0
Bleeding varicose vein (Vascular disorders) | 0 | 2
Blood pressure inadequately controlled (Vascular disorders) | 0 | 1
Circulatory collapse (Vascular disorders) | 5 | 8
Deep vein thrombosis (Vascular disorders) | 5 | 5
Diabetic vascular disorder (Vascular disorders) | 1 | 0
Extremity necrosis (Vascular disorders) | 2 | 0
Femoral artery embolism (Vascular disorders) | 0 | 1
Femoral artery occlusion (Vascular disorders) | 3 | 6
Haematoma (Vascular disorders) | 2 | 1
Haemorrhage (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 13 | 12
Hypertensive crisis (Vascular disorders) | 7 | 2
Hypertensive emergency (Vascular disorders) | 0 | 2
Hypoperfusion (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 59 | 68
Hypovolaemic shock (Vascular disorders) | 5 | 2
Iliac artery occlusion (Vascular disorders) | 0 | 3
Intermittent claudication (Vascular disorders) | 2 | 3
Ischaemia (Vascular disorders) | 0 | 1
Jugular vein thrombosis (Vascular disorders) | 1 | 0
Lymphatic fistula (Vascular disorders) | 0 | 1
Lymphocele (Vascular disorders) | 1 | 0
Lymphoedema (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 5 | 3
Peripheral arterial occlusive disease (Vascular disorders) | 22 | 13
Peripheral artery aneurysm (Vascular disorders) | 3 | 1
Peripheral artery stenosis (Vascular disorders) | 4 | 2
Peripheral artery thrombosis (Vascular disorders) | 4 | 3
Peripheral circulatory failure (Vascular disorders) | 1 | 0
Peripheral embolism (Vascular disorders) | 4 | 2
Peripheral ischaemia (Vascular disorders) | 18 | 8
Peripheral vascular disorder (Vascular disorders) | 7 | 5
Phlebitis (Vascular disorders) | 2 | 0
Polyarteritis nodosa (Vascular disorders) | 0 | 1
Shock (Vascular disorders) | 4 | 5
Shock haemorrhagic (Vascular disorders) | 0 | 1
Subgaleal haematoma (Vascular disorders) | 0 | 1
Superior vena cava syndrome (Vascular disorders) | 0 | 1
Thrombophlebitis (Vascular disorders) | 3 | 3
Thrombophlebitis superficial (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 1 | 2
Varicose vein (Vascular disorders) | 0 | 2
Vascular compression (Vascular disorders) | 1 | 0
Vasculitis (Vascular disorders) | 2 | 0
Vein collapse (Vascular disorders) | 1 | 0
Venous haemorrhage (Vascular disorders) | 0 | 1
Venous insufficiency (Vascular disorders) | 0 | 3
Venous thrombosis (Vascular disorders) | 0 | 1
Venous thrombosis limb (Vascular disorders) | 1 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LCZ696 (N=4203) | Enalapril (N=4229)
Anaemia (Blood and lymphatic system disorders) | 140 | 160
Angina pectoris (Cardiac disorders) | 125 | 125
Atrial fibrillation (Cardiac disorders) | 159 | 137
Cardiac failure (Cardiac disorders) | 214 | 274
Constipation (Gastrointestinal disorders) | 85 | 120
Diarrhoea (Gastrointestinal disorders) | 175 | 179
Nausea (Gastrointestinal disorders) | 82 | 96
Fatigue (General disorders) | 124 | 121
Non-cardiac chest pain (General disorders) | 77 | 92
Oedema peripheral (General disorders) | 205 | 201
Bronchitis (Infections and infestations) | 166 | 202
Influenza (Infections and infestations) | 154 | 128
Nasopharyngitis (Infections and infestations) | 204 | 174
Pneumonia (Infections and infestations) | 91 | 70
Upper respiratory tract infection (Infections and infestations) | 199 | 191
Urinary tract infection (Infections and infestations) | 166 | 167
Diabetes mellitus (Metabolism and nutrition disorders) | 101 | 112
Gout (Metabolism and nutrition disorders) | 116 | 114
Hyperkalaemia (Metabolism and nutrition disorders) | 477 | 569
Hyperuricaemia (Metabolism and nutrition disorders) | 108 | 149
Hypokalaemia (Metabolism and nutrition disorders) | 130 | 98
Arthralgia (Musculoskeletal and connective tissue disorders) | 124 | 117
Back pain (Musculoskeletal and connective tissue disorders) | 157 | 138
Pain in extremity (Musculoskeletal and connective tissue disorders) | 91 | 98
Dizziness (Nervous system disorders) | 259 | 202
Headache (Nervous system disorders) | 100 | 106
Insomnia (Psychiatric disorders) | 92 | 91
Renal failure (Renal and urinary disorders) | 73 | 97
Renal impairment (Renal and urinary disorders) | 393 | 449
Cough (Respiratory, thoracic and mediastinal disorders) | 367 | 528
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 173 | 263
Hypertension (Vascular disorders) | 115 | 185
Hypotension (Vascular disorders) | 700 | 454

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.